CLINICAL TRIAL: NCT02308163
Title: Phase 3 Study of ASP015K - A Randomized, Double-blind, Placebo-controlled Confirmatory Study of the Safety and Efficacy of ASP015K in Patients With Rheumatoid Arthritis Who Had an Inadequate Response to DMARDs
Brief Title: A Study to Evaluate Safety and Efficacy of ASP015K in Patients With Rheumatoid Arthritis (RA) Who Had an Inadequate Response to DMARDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015K-CL-RAJ3
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; ASP015K
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants were assigned to receive placebo to peficitinib once a day until week 12.
  Interventions: Drug: Placebo
- Peficitinib 100 mg (Experimental): Participants were assigned to receive peficitinib 100 mg/day for 52 weeks.
  Interventions: Drug: Peficitinib
- Peficitinib 150 mg (Experimental): Participants were assigned to receive peficitinib 150 mg/day for 52 weeks.
  Interventions: Drug: Peficitinib
- Etanercept (Active Comparator): Participants were administered 50 mg of subcutaneous etanercept once weekly for 52 weeks.
  Interventions: Biological: Etanercept

INTERVENTIONS:
Drug: Peficitinib — oral
  Other Names: ASP015K
  Arms: Peficitinib 100 mg; Peficitinib 150 mg
Drug: Placebo — oral
  Arms: Placebo
Biological: Etanercept — subcutaneous injection
  Arms: Etanercept

SUMMARY:
The objective of this study was to verify the superiority of ASP015K alone or in combination with disease-modifying antirheumatic drugs (DMARDs) over placebo in terms of efficacy in participants with rheumatoid arthritis (RA) who had an inadequate response to DMARDs

DETAILED DESCRIPTION:
This was a multi-center, randomized, placebo-controlled, double-blind, parallel-group, confirmatory study to evaluate the efficacy and safety of ASP015K alone or in combination with DMARDs in participants with RA who had an inadequate response to DMARDs.

Etanercept was also administered as the reference drug in an open-label manner. The study drug was orally administered once daily (QD) after breakfast for 52 weeks. Etanercept was administered subcutaneously QD for 52 weeks. At Week 12, participants in the placebo group were switched to ASP015K.

The dose of ASP015K to be started at Week 12 for the placebo group was determined randomly at baseline in advance and switched in a blinded manner.

Participants in ASP015K group or placebo groups who had completed the study were eligible for participation in an open-label extension study (015K-CL-RAJ2).

ELIGIBILITY:
Inclusion Criteria:

* Subject has RA diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria
* Subject who did not receive the following drugs, or received the drugs with stable dosage for at least 28 days prior to the baseline (start of treatment) for RA treatment:

  * Non-steroidal anti-inflammatory drugs (NSAIDs; excluding topical formulations), oral morphine or equivalent opioid analgesics (≤ 30 mg/day), acetaminophen, or oral corticosteroids (≤ 10 mg/day in prednisolone equivalent)
* At screening subject has active RA as evidenced by both of the following:

  * ≥ 6 tender/painful joints (using 68-joint assessment)
  * ≥ 6 swollen joints (using 66-joint assessment)
* CRP > 0.50 mg/dL at screening
* Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class I, II or, III at screening.
* Inadequate responder to (including subjects who were intolerant of) at least one DMARD administered for at least 90 days prior to screening

Exclusion Criteria:

* Subject has received a biologic DMARD within the specified period
* Subject has received etanercept
* Inadequate responder to at least 3 biologic DMARDs as determined by investigator/sub-investigator
* Subject has received intra-articular, intravenous, intramuscular or endorectal (excluding suppositories for anal diseases) corticosteroid within 28 days prior to baseline
* Subject has participated in any study of ASP015K and has received ASP015K or placebo
* Subject has received other investigational drugs within 90 days or within 5 half-lives, whichever is longer, prior to baseline
* Subject has received plasma exchange therapy within 60 days prior to baseline
* Subject has undergone joint drainage, has received local anesthesia and nerve block, or has received articular cartilage protectant at the assessed joint within 28 days prior to baseline
* Subject has undergone surgery and has residual effects in the assessed joints at the discretion of investigator/sub-investigator, or is scheduled to undergo surgery that may affect the study evaluation of the assessed joints at the discretion of investigator/sub-investigator
* A diagnosis of inflammatory arthritis (psoriatic arthritis, ankylosing spondylitis, SLE, sarcoidosis, etc.) other than RA
* Any of the following laboratory values at screening:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count < 1000/μL
  * Absolute lymphocyte count < 800/μL
  * Platelet count < 75000/μL
  * ALT ≥ 2 ×ULN
  * AST ≥ 2 × ULN
  * Total bilirubin (TBL) ≥ 1.5 × ULN
  * Estimated GFR ≤ 40 mL/min as measured by the MDRD method
  * β-D-glucan > ULN [in case of Japan: ≥ 11 pg/mL]
  * Positive HBs antigen, HBc antibody, HBs antibody or HBV-DNA quantitation (However, subject with negative HBs antigen and HBV-DNA quantitation, and positive HBc antibody and/or HBs antibody is eligible if HBV-DNA is monitored by HBV-DNA quantitation at every scheduled visit after initiation of study drug or reference drug administration.)
  * Positive HCV antibody
* Subject has a history of or concurrent active tuberculosis (TB)
* Subject has a history of or concurrent interstitial pneumonia and investigator/sub-investigator judges that it is inappropriate for the subject to participate in this study
* Subject has a history of or concurrent malignant tumor (except for successfully treated basal cell carcinoma)
* Subject has received live or live attenuated virus vaccination within 56 days prior to baseline. (Inactivated vaccines including influenza and pneumococcal vaccines are allowed.)
* Subject has a history of or concurrent demyelinating disorders
* Subject has any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, infectious, or autoimmune disease except for RA (excluding Sjogren's syndrome and chronic thyroiditis), or any ongoing illness which would make the subject unsuitable for the study as determined by the investigator/sub-investigator
* Subject has a history of clinically significant allergy. (Clinically significant allergy includes allergies such as systemic urticaria induced by specific antigens and drugs, anaphylaxis, and allergy associated with shock necessitating hospitalized treatment.)
* Subject has concurrent cardiac failure, defined as NYHA classification Class III or higher, or a history of it
* Subject has concurrent prolonged QT syndrome or a history of it. Subject has prolonged QT interval (defined as QTc ≥ 500 msec. Subject has QTc ≥ 500 msec at retest will be excluded) at screening
* Subject has a history of positive HIV infection
* Subject has congenital short QT syndrome or a history of it. Subject has shortened QT interval (defined as QTc < 330 msec. Subject has QTc < 330 msec at retest will be excluded) at screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (153):
- Japan (132):
  - JP00037, Nagoya, Aichi-ken
  - JP00109, Nagoya, Aichi-ken
  - JP00130, Nagoya, Aichi-ken
  - JP00066, Okazaki, Aichi-ken
  - JP00140, Toyoake, Aichi-ken
  - JP00108, Toyohashi, Aichi-ken
  - JP00156, Toyota, Aichi-ken
  - JP00068, Yatomi, Aichi-ken
  - JP00102, Kamagaya, Chiba
  - JP00127, Matsudo, Chiba
  - JP00115, Narashino, Chiba
  - JP00138, Yotsukaidō, Chiba
  - JP00120, Iizuka, Fukuoka
  - JP00040, Kitakyushu, Fukuoka
  - JP00119, Kitakyushu, Fukuoka
  - JP00071, Kurume, Fukuoka
  - JP00097, Kurume, Fukuoka
  - JP00106, Kurume, Fukuoka
  - JP00033, Takasaki, Gunma
  - JP00026, Asahikawa, Hokkaido
  - JP00090, Hakodate, Hokkaido
  - JP00125, Kushiro, Hokkaido
  - JP00001, Sapporo, Hokkaido
  - JP00002, Sapporo, Hokkaido
  - JP00003, Sapporo, Hokkaido
  - JP00031, Sapporo, Hokkaido
  - JP00038, Sapporo, Hokkaido
  - JP00114, Sapporo, Hokkaido
  - JP00158, Sapporo, Hokkaido
  - JP00056, Akashi, Hyōgo
  - JP00069, Himeji, Hyōgo
  - JP00113, Kakogawa, Hyōgo
  - JP00041, Katō, Hyōgo
  - JP00042, Kobe, Hyōgo
  - JP00092, Kobe, Hyōgo
  - JP00154, Kobe, Hyōgo
  - JP00117, Nishinomiya, Hyōgo
  - JP00107, Hitachi, Ibaraki
  - JP00073, Koga, Ibaraki
  - JP00054, Mito, Ibaraki
  - JP00049, Morioka, Iwate
  - JP00084, Isehara, Kanagawa
  - JP00048, Kawasaki, Kanagawa
  - JP00058, Kawasaki, Kanagawa
  - JP00141, Sagamihara, Kanagawa
  - JP00096, Yokohama, Kanagawa
  - JP00128, Yokosuka, Kanagawa
  - JP00057, Tamana, Kumamoto
  - JP00004, Sendai, Miyagi
  - JP00027, Sendai, Miyagi
  - JP00036, Sendai, Miyagi
  - JP00105, Sendai, Miyagi
  - JP00151, Sendai, Miyagi
  - JP00050, Hyūga, Miyazaki
  - JP00162, Isehaya, Nagasaki
  - JP00101, Ōmura, Nagasaki
  - JP00103, Ōmura, Nagasaki
  - JP00153, Sasebo, Nagasaki
  - JP00094, Kashihara, Nara
  - JP00025, Nagaoka, Niigata
  - JP00144, Shibata, Niigata
  - JP00064, Beppu, Oita Prefecture
  - JP00051, Setouchi, Okayama-ken
  - JP00011, Hannan, Osaka
  - JP00134, Higashiosaka, Osaka
  - JP00078, Kawachi-Nagano, Osaka
  - JP00137, Sakai, Osaka
  - JP00070, Suita, Osaka
  - JP00086, Suita, Osaka
  - JP00061, Toyonaka, Osaka
  - JP00075, Ureshino, Saga-ken
  - JP00126, Gyōda, Saitama
  - JP00007, Hiki, Saitama
  - JP00082, Iruma, Saitama
  - JP00060, Kawagoe, Saitama
  - JP00161, Kawagoe, Saitama
  - JP00062, Kawaguchi, Saitama
  - JP00052, Sayama, Saitama
  - JP00008, Tokorozawa, Saitama
  - JP00133, Kakegawa, Shizuoka
  - JP00077, Kanuma, Tochigi
  - JP00024, Bunkyo, Tokyo
  - JP00043, Bunkyo, Tokyo
  - JP00149, Bunkyo, Tokyo
  - JP00152, Bunkyo, Tokyo
  - JP00095, Chiyoda City, Tokyo
  - JP00099, Chiyoda City, Tokyo
  - JP00142, Chūō, Tokyo
  - JP00063, Hachiōji, Tokyo
  - JP00053, Kiyose, Tokyo
  - JP00072, Meguro City, Tokyo
  - JP00083, Meguro City, Tokyo
  - JP00148, Ōta-ku, Tokyo
  - JP00100, Setagaya City, Tokyo
  - JP00032, Shinjuku, Tokyo
  - JP00010, Takaoka, Toyama
  - JP00155, Nishimuro, Wakayama
  - JP00104, Shimonoseki, Yamaguchi
  - JP00047, Shūnan, Yamaguchi
  - JP00018, Fukuoka
  - JP00020, Fukuoka
  - JP00035, Fukuoka
  - JP00059, Fukuoka
  - JP00067, Fukuoka
  - JP00076, Fukuoka
  - JP00131, Fukuoka
  - JP00164, Fukuoka
  - JP00013, Hiroshima
  - JP00014, Hiroshima
  - JP00015, Hiroshima
  - JP00016, Hiroshima
  - JP00055, Hiroshima
  - JP00065, Kagoshima
  - JP00074, Kagoshima
  - JP00093, Kochi
  - JP00022, Kumamoto
  - JP00046, Kumamoto
  - JP00123, Kyoto
  - JP00159, Kyoto
  - JP00023, Miyagi
  - JP00122, Miyazaki
  - JP00080, Nagano
  - JP00098, Nagasaki
  - JP00112, Nagasaki
  - JP00147, Nagasaki
  - JP00118, Okayama
  - JP00150, Osaka
  - JP00157, Osaka
  - JP00017, Ōita
  - JP00089, Shizuoka
  - JP00135, Shizuoka
  - JP00139, Toyama
- South Korea (11):
  - KR00504, Daegu
  - KR00510, Daegu
  - KR00505, Gwangju
  - KR00506, Incheon
  - KR00508, Jeonju
  - KR00501, Seoul
  - KR00502, Seoul
  - KR00503, Seoul
  - KR00509, Seoul
  - KR00511, Seoul
  - KR00507, Suwon
- Taiwan (10):
  - TW00708, Kaohsiung City
  - TW00709, Kaohsiung City
  - TW00704, Taichung
  - TW00705, Taichung
  - TW00710, Taichung
  - TW00712, Tainan
  - TW00701, Taipei
  - TW00702, Taipei
  - TW00711, Taipei
  - TW00703, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Tanaka Y, Takeuchi T, Izutsu H, Kaneko Y, Kato D, Fukuda M, Rokuda M, Schultz NM. Patient- and physician-reported outcomes from two phase 3 randomized studies (RAJ3 and RAJ4) of peficitinib (ASP015K) in Asian patients with rheumatoid arthritis. Arthritis Res Ther. 2021 Aug 24;23(1):221. doi: 10.1186/s13075-021-02590-z. PMID 34429152
- [Derived] Toyoshima J, Kaibara A, Shibata M, Kaneko Y, Izutsu H, Nishimura T. Exposure-response modeling of peficitinib efficacy in patients with rheumatoid arthritis. Pharmacol Res Perspect. 2021 May;9(3):e00744. doi: 10.1002/prp2.744. PMID 33929089
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028
- [Derived] Tanaka Y, Takeuchi T, Tanaka S, Kawakami A, Iwasaki M, Song YW, Chen YH, Wei JC, Lee SH, Rokuda M, Izutsu H, Ushijima S, Kaneko Y, Akazawa R, Shiomi T, Yamada E. Efficacy and safety of peficitinib (ASP015K) in patients with rheumatoid arthritis and an inadequate response to conventional DMARDs: a randomised, double-blind, placebo-controlled phase III trial (RAJ3). Ann Rheum Dis. 2019 Oct;78(10):1320-1332. doi: 10.1136/annrheumdis-2019-215163. Epub 2019 Jul 26. PMID 31350270
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with rheumatoid arthritis (RA) who had an inadequate response to disease-modifying antirheumatic drugs (DMARDs) were enrolled in 142 sites in Japan, 11 sites in Korea and 12 sites in Taiwan.
Pre-assignment Details: Participants were randomized in a 1:1:1:2 ratio to peficitinib 100 mg, 150 mg, placebo or etanercept groups at baseline. At week 12, participants in the placebo group were switched to receive either peficitinib at a dose of 100 mg or 150 mg. The dose of peficitinib administered to the placebo group from week 12 was determined in advance randomly.
Groups:
- Placebo / Peficitinib 100 mg: Participants were assigned to receive placebo to peficitinib once a day until week 12 and peficitinib 100 mg/day from week 12 to week 52.
- Placebo / Peficitinib 150 mg: Participants were assigned to receive placebo to peficitinib once a day until week 12 and peficitinib 150 mg/day from week 12 to week 52.
Period: Overall Study
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Started | 104 | 102 | 50 | 52 | 201
Completed | 73 | 84 | 36 | 39 | 167
Not Completed | 31 | 18 | 14 | 13 | 34
Not completed — Not fulfill eligible criteria | 1 | 2 | 0 | 1 | 1
Not completed — Adverse Event | 9 | 5 | 2 | 2 | 11
Not completed — Lack of Efficacy | 11 | 3 | 8 | 4 | 6
Not completed — Withdrawal of consent | 2 | 3 | 0 | 2 | 6
Not completed — Protocol Violation | 3 | 3 | 3 | 2 | 5
Not completed — Lab data met discontinuation criteria | 3 | 0 | 0 | 2 | 0
Not completed — Miscellaneous | 2 | 2 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) was defined as all participants who received at least 1 dose of the study drug or reference drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept | Placebo | Total
Number analyzed (Participants) | 104 | 102 | 200 | 101 | 507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (12.2) | 55 (12.8) | 55.5 (11.6) | 56.3 (11.7) | 55.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 78 | 138 | 73 | 366
  Male | 27 | 24 | 62 | 28 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 104 | 102 | 200 | 101 | 507
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Tender Joint Count (68 Joints) [Mean (Standard Deviation); unit: tender joints] — Population: The full analysis set (FAS) consisted of all participants who were randomized and received at least 1 dose of the study drug or reference drug.
  tender joints | 15 (9.4) | 15.4 (9.5) | 14.9 (9.3) | 16.2 (10.7) | 15.3 (9.6)
Swollen Joint Count (66 Joints) [Mean (Standard Deviation); unit: swollen joints] — Population: FAS
  swollen joints | 12.4 (6.3) | 12.8 (7.1) | 11.9 (6.8) | 12.9 (7.2) | 12.4 (6.8)
Subject's Global Assessment of Arthritis Pain [Mean (Standard Deviation); unit: units on a scale] — The participants assessed his/her own pain severity on a Visual analog scale (VAS) from 0-100 mm on the questionnaire form. Higher scores indicated greater activity pain. Population: FAS
  units on a scale | 57.31 (26.71) | 58.02 (25.66) | 55.79 (26.54) | 57.56 (25.07) | 56.9 (26.05)
Subject's Global Assessment of Arthritis [Mean (Standard Deviation); unit: units on a scale] — The participants assessed his/her own disease activity on a VAS of 0-100 mm on the questionnaire form. Higher scores indicated greater activity impairment. Population: FAS
  units on a scale | 57.54 (24.78) | 59.52 (25.73) | 57.52 (26.92) | 58.99 (25.7) | 58.22 (25.95)
Physician's Global Assessment of Arthritis [Mean (Standard Deviation); unit: units on a scale] — The investigator assessed the participants' disease activity on a VAS of 0-100 mm on the physician assessment table. Higher scores indicated greater activity impairment. Population: FAS
  units on a scale | 60.21 (20.11) | 58.46 (19.35) | 58.17 (19.87) | 61.93 (19.35) | 59.39 (19.71)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI (range 0 - 3) was composed of 20 items in 8 categories (Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, and Activities). Each category had at least two questions. Within each category, participants reported the amount of difficulty they had in performing the specific question items. Higher HAQ-DI score indicated greater disease activity. Population: FAS
  units on a scale | 0.92 (0.69) | 1.03 (0.67) | 1.03 (0.75) | 1 (0.66) | 1 (0.7)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dL] — Population: FAS
  mg/dL | 2.296 (2.566) | 2.561 (2.597) | 2.055 (2.144) | 2.258 (2.224) | 2.247 (2.346)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: mm/h] — Population: FAS
  mm/h | 49.6 (27.4) | 50.6 (29.7) | 47.4 (29.8) | 47.9 (27.6) | 48.6 (28.8)
Prior Biologic Disease-modifying Antirheumatic Drug-inadequate Response (DMARD-IR) [Count of Participants; unit: Participants] — For the participants whose "Reactivity" was selected as "Inadequate Response" or "Unknown", "Prior Biologic DMARD-IR" was regarded as "Yes", Otherwise "No". Population: FAS
  Participants
    No | 95 | 95 | 185 | 96 | 471
    Yes | 9 | 7 | 15 | 5 | 36
Concomitant DMARD at Baseline [Count of Participants; unit: Participants] — Concomitant DMARD at Baseline used at the initiation of treatment with the study drug or reference drug was regarded as "Yes", Otherwise "No". Population: FAS
  Participants
    No | 13 | 13 | 24 | 14 | 64
    Yes | 91 | 89 | 176 | 87 | 443
Study Region [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Japan | 85 | 83 | 164 | 83 | 415
    Korea | 11 | 11 | 22 | 10 | 54
    Taiwan | 8 | 8 | 14 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) C-Reactive Protein (CRP) Response at Week 12
Description: The ACR20 response required that all criteria from (1) to (3) below be met.
  1. Tender joint count (TJC) : ≥ 20% reduction compared with baseline.
  2. Swollen joint count (SJC) : ≥ 20% reduction compared with baseline.
  3. ≥ 20% improvement in 3 or more of the following 5 parameters compared with baseline
  (3) ≥ 20% improvement in 3 or more of the following 5 parameters compared with baseline: Subject's assessment of pain, Subject's Global Assessment of Arthritis (SGA), Physician's Global Assessment of Arthritis (PGA), Health Assessment Questionnaire - Disability Index (HAQ-DI), C-Reactive Protein (CRP).
Time Frame: Baseline and Week 12/early termination (ET)
Population: The analysis population consisted of the Full Analysis Set (FAS). Last observation carried forward (LOCF) was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 101 | 104 | 102 | 200
Percentage of Participants | 30.7 | 57.7 | 74.5 | 83.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — Closed testing procedure was used for multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 3.13, 95% CI 2-sided [1.76 to 5.58] — Based on logistic regression model: ACR20-CRP response (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 6.59, 95% CI 2-sided [3.56 to 12.20] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With an ACR20-CRP Response Through Week 52
Description: The ACR20 response required that all criteria from (1) to (3) below be met.
  1. TJC : ≥ 20% reduction compared with baseline.
  2. SJC : ≥ 20% reduction compared with baseline.
  3. ≥ 20% improvement in 3 or more of the following 5 parameters compared with baseline: Subject's assessment of pain, SGA, PGA, HAQ-DI, CRP.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | 43.9 | 45.0 | 21.4 | 19.1 | 61.0
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | 51.0 | 68.7 | 38.1 | 25.5 | 80.5
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | 59.4 | 77.2 | 31.7 | 34.0 | 84.8
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | 64.5 | 79.6 | 58.5 | 61.7 | 86.7
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | 64.1 | 81.5 | 51.2 | 71.7 | 88.5
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | 63.2 | 85.6 | 61.5 | 71.1 | 90.1
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | 72.3 | 87.6 | 60.0 | 67.4 | 92.7
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | 76.5 | 88.4 | 63.9 | 73.3 | 88.1
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | 72.2 | 90.7 | 66.7 | 76.7 | 92.0
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | 73.7 | 90.7 | 67.6 | 83.3 | 92.5
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 74.7 | 88.2 | 79.4 | 84.6 | 91.2
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | 74.3 | 90.5 | 73.5 | 82.1 | 90.5
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 73.2 | 90.1 | 79.4 | 81.6 | 90.7
  End of Treatment (EOT) | 65.4 | 84.3 | 67.4 | 74.5 | 86.5

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50)-CRP Response at Week 12
Description: The ACR50 response required that all criteria from (1) to (3) below be met.
  1. TJC : ≥ 50% reduction compared with baseline.
  2. SJC : ≥ 50% reduction compared with baseline.
  3. ≥ 50% improvement in 3 or more of the following 5 parameters compared with baseline: Subject's assessment of pain, SGA, PGA, HAQ-DI, CRP.
Time Frame: Baseline and Week 12/ET
Population: FAS. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 101 | 104 | 102 | 200
Percentage of Participants | 8.9 | 30.8 | 42.2 | 52.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 4.79, 95% CI 2-sided [2.14 to 10.75] — Based on logistic regression model: ACR50-CRP response (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 7.86, 95% CI 2-sided [3.53 to 17.50] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants With an ACR50-CRP Response Through Week 52
Description: as for outcome 3
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | 8.2 | 14.0 | 4.8 | 2.1 | 29.5
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | 25.0 | 35.4 | 4.8 | 6.4 | 47.2
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | 32.3 | 45.7 | 7.3 | 12.8 | 55.0
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | 43.0 | 45.2 | 31.7 | 25.5 | 60.6
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | 41.3 | 54.3 | 22.0 | 43.5 | 66.5
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | 43.7 | 62.2 | 38.5 | 44.4 | 64.8
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | 44.6 | 60.7 | 40.0 | 50.0 | 69.5
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | 50.6 | 65.1 | 52.8 | 44.4 | 70.5
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | 53.2 | 68.6 | 47.2 | 44.2 | 70.3
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | 47.4 | 69.8 | 45.9 | 52.4 | 73.4
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 50.7 | 69.4 | 50.0 | 53.8 | 70.2
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | 48.6 | 73.8 | 58.8 | 69.2 | 75.6
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 49.3 | 75.3 | 47.1 | 65.8 | 77.2
  EOT | 43.3 | 66.7 | 41.9 | 55.3 | 69.0

5. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70)-CRP Response at Week 12
Description: The ACR70 response required that all criteria from (1) to (3) below be met.
  1. TJC : ≥ 70% reduction compared with baseline.
  2. SJC : ≥ 70% reduction compared with baseline.
  3. ≥ 70% improvement in 3 or more of the following 5 parameters compared with baseline: Subject's assessment of pain, SGA, PGA, HAQ-DI, CRP.
Time Frame: Baseline and Week 12/ET
Population: FAS. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 101 | 104 | 102 | 200
Percentage of Participants | 1.0 | 13.5 | 27.5 | 30.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo. Difference vs. Peficitinib 100mg was not estimable; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 39.93, 95% CI 2-sided [5.29 to 301.61] — Based on logistic regression model: ACR70-CRP response (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)

6. Secondary Outcome: Percentage of Participants With an ACR70-CRP Response Through Week 52
Description: as for outcome 5
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | 1.0 | 2.0 | 0.0 | 0.0 | 14.5
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | 11.5 | 14.1 | 0.0 | 2.1 | 20.5
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | 14.6 | 29.3 | 0.0 | 2.1 | 31.9
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | 23.7 | 28.0 | 7.3 | 8.5 | 37.8
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | 26.1 | 30.4 | 7.3 | 19.6 | 41.8
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | 28.7 | 40.0 | 15.4 | 22.2 | 44.5
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | 25.3 | 38.2 | 20.0 | 17.4 | 48.0
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | 28.4 | 39.5 | 25.0 | 24.4 | 47.7
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | 31.6 | 43.0 | 27.8 | 18.6 | 44.6
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | 28.9 | 47.7 | 27.0 | 35.7 | 49.7
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 30.7 | 49.4 | 41.2 | 28.2 | 52.0
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | 33.8 | 51.2 | 32.4 | 38.5 | 54.2
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 35.2 | 48.1 | 38.2 | 42.1 | 56.2
  EOT | 31.7 | 42.2 | 34.9 | 34.0 | 48.0

7. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) 28-CRP at Week 12
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to below description.
  DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. Higher DAS28 score indicated greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 101 | 101 | 200
Units on a Scale | -0.64 (1.20) | -1.62 (1.41) | -2.17 (1.14) | -2.42 (1.11)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -1.06, 95% CI 2-sided [-1.41 to -0.71], Standard Error of Mean 0.18 — Based on analysis of covariance model: DAS28 Change = Treatment + Baseline DAS28 + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -1.55, 95% CI 2-sided [-1.86 to -1.24], Standard Error of Mean 0.16 — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline DAS28-CRP Through Week 52
Description: as for outcome 7
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -1.11 (0.97) | -1.29 (0.83) | -0.49 (0.78) | -0.56 (0.86) | -1.89 (1.05)
  Week 8: number analyzed (Participants) | 96 | 98 | 42 | 47 | 195
  Week 8 | -1.48 (1.24) | -1.92 (0.96) | -0.70 (1.02) | -0.65 (1.00) | -2.27 (1.03)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -1.66 (1.34) | -2.27 (1.12) | -0.70 (1.23) | -0.82 (1.15) | -2.49 (1.06)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -1.96 (1.37) | -2.40 (1.26) | -1.60 (1.29) | -1.92 (1.25) | -2.61 (1.01)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -2.01 (1.41) | -2.57 (1.20) | -1.58 (1.42) | -2.15 (1.22) | -2.73 (1.04)
  Week 24: number analyzed (Participants) | 87 | 89 | 39 | 45 | 182
  Week 24 | -2.06 (1.39) | -2.68 (1.24) | -1.60 (1.34) | -2.28 (1.30) | -2.79 (1.04)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -2.12 (1.37) | -2.80 (1.27) | -1.90 (1.50) | -2.35 (1.31) | -2.90 (0.97)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -2.26 (1.30) | -2.77 (1.29) | -1.98 (1.47) | -2.22 (1.35) | -2.94 (1.05)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -2.31 (1.34) | -2.87 (1.22) | -2.21 (1.40) | -2.26 (1.35) | -2.91 (1.03)
  Week 40: number analyzed (Participants) | 75 | 86 | 37 | 42 | 173
  Week 40 | -2.31 (1.36) | -2.88 (1.27) | -2.17 (1.46) | -2.47 (1.48) | -2.99 (0.97)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -2.34 (1.29) | -2.86 (1.37) | -2.39 (1.35) | -2.47 (1.42) | -2.97 (0.95)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -2.26 (1.31) | -2.98 (1.27) | -2.58 (1.32) | -2.73 (1.29) | -3.03 (1.01)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -2.28 (1.38) | -2.99 (1.26) | -2.51 (1.29) | -2.73 (1.30) | -3.04 (1.08)
  EOT: number analyzed (Participants) | 101 | 101 | 42 | 47 | 200
  EOT | -2.01 (1.63) | -2.75 (1.36) | -2.11 (1.59) | -2.50 (1.41) | -2.80 (1.19)

9. Secondary Outcome: Change From Baseline in DAS28-Erythrocyte Sedimentation Rate (ESR) at Week 12
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to below description.
  DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. Higher DAS28 score indicated greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 98 | 102 | 101 | 198
Units on a Scale | -0.62 (1.17) | -1.60 (1.39) | -2.24 (1.23) | -2.51 (1.27)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -1.03, 95% CI 2-sided [-1.38 to -0.67], Standard Error of Mean 0.18 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -1.64, 95% CI 2-sided [-1.96 to -1.31], Standard Error of Mean 0.17 — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in DAS28-ESR Through Week 52
Description: as for outcome 9
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 46 | 199
  Week 4 | -1.13 (0.94) | -1.26 (0.84) | -0.46 (0.74) | -0.63 (0.87) | -1.90 (1.12)
  Week 8: number analyzed (Participants) | 95 | 98 | 42 | 45 | 194
  Week 8 | -1.50 (1.20) | -1.96 (1.04) | -0.68 (0.99) | -0.57 (0.92) | -2.33 (1.12)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 46 | 190
  Week 12 | -1.65 (1.33) | -2.35 (1.21) | -0.66 (1.18) | -0.80 (1.13) | -2.58 (1.22)
  Week 16: number analyzed (Participants) | 93 | 92 | 41 | 46 | 188
  Week 16 | -1.95 (1.40) | -2.50 (1.36) | -1.53 (1.33) | -1.84 (1.20) | -2.68 (1.15)
  Week 20: number analyzed (Participants) | 91 | 91 | 40 | 45 | 181
  Week 20 | -2.06 (1.44) | -2.65 (1.29) | -1.57 (1.43) | -2.15 (1.20) | -2.76 (1.15)
  Week 24: number analyzed (Participants) | 87 | 88 | 38 | 44 | 181
  Week 24 | -2.11 (1.47) | -2.79 (1.39) | -1.60 (1.37) | -2.25 (1.16) | -2.86 (1.18)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 45 | 176
  Week 28 | -2.14 (1.43) | -2.87 (1.37) | -1.94 (1.51) | -2.31 (1.29) | -2.97 (1.14)
  Week 32: number analyzed (Participants) | 81 | 86 | 35 | 44 | 175
  Week 32 | -2.28 (1.41) | -2.88 (1.41) | -1.98 (1.46) | -2.26 (1.44) | -3.01 (1.13)
  Week 36: number analyzed (Participants) | 79 | 85 | 35 | 42 | 175
  Week 36 | -2.38 (1.43) | -3.00 (1.36) | -2.18 (1.39) | -2.28 (1.35) | -3.00 (1.14)
  Week 40: number analyzed (Participants) | 76 | 86 | 36 | 41 | 173
  Week 40 | -2.38 (1.44) | -3.02 (1.38) | -2.12 (1.44) | -2.49 (1.60) | -3.10 (1.06)
  Week 44: number analyzed (Participants) | 75 | 85 | 33 | 39 | 171
  Week 44 | -2.40 (1.39) | -3.02 (1.51) | -2.39 (1.34) | -2.55 (1.38) | -3.05 (1.04)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 38 | 168
  Week 48 | -2.32 (1.40) | -3.09 (1.44) | -2.67 (1.39) | -2.79 (1.28) | -3.16 (1.09)
  Week 52: number analyzed (Participants) | 71 | 81 | 33 | 37 | 162
  Week 52 | -2.35 (1.48) | -3.06 (1.40) | -2.45 (1.30) | -2.67 (1.23) | -3.10 (1.16)
  EOT: number analyzed (Participants) | 102 | 101 | 41 | 46 | 199
  EOT | -2.06 (1.70) | -2.81 (1.47) | -2.06 (1.56) | -2.44 (1.44) | -2.86 (1.27)

11. Secondary Outcome: Change From Baseline in TJC (68 Joints) at Week 12
Description: The following 68 joints subjects to assessment were examined for tender joints and the location was confirmed. Higher TJC68 indicated greater disease activity.
  Temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2), elbow joints (2), wrist joints (2), distal interphalangeal joints (8), proximal interphalangeal joints of both hands (10), metacarpophalangeal joints (10), hip joints (2), knee joints (2), ankle joints (2), tarsal bones (2), metatarsophalangeal joints (10), interphalangeal joint joints of toes (2), proximal interphalangeal joints of both feet (8).
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Tender Joints | -4.3 (9.2) | -8.2 (8.8) | -9.9 (8.0) | -10.7 (7.8)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -4.6, 95% CI 2-sided [-6.8 to -2.4], Standard Error of Mean 1.1 — Based on analysis of covariance model: TJC68 Change = Treatment + Baseline TJC68 + the prior biologic - DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -6.1, 95% CI 2-sided [-8.1 to -4.0], Standard Error of Mean 1.0 — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in TJC (68 Joints) Through Week 52
Description: as for outcome 11
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Tender Joints
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -5.9 (8.0) | -5.4 (6.0) | -3.9 (8.1) | -4.3 (6.4) | -8.3 (7.7)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -7.8 (7.6) | -8.6 (7.1) | -4.4 (8.4) | -3.9 (8.3) | -10.3 (7.1)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -8.6 (8.8) | -10.3 (8.0) | -5.0 (9.7) | -5.5 (7.6) | -11.0 (7.6)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -9.2 (9.2) | -10.3 (8.8) | -7.7 (10.2) | -9.6 (7.5) | -11.5 (7.6)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -9.8 (9.2) | -11.3 (8.6) | -8.1 (10.8) | -10.3 (7.9) | -12.0 (7.9)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 46 | 182
  Week 24 | -9.4 (9.4) | -11.3 (9.7) | -7.6 (9.9) | -11.7 (7.9) | -12.2 (8.2)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -9.7 (8.8) | -12.0 (9.3) | -8.4 (10.3) | -11.5 (8.2) | -12.6 (8.6)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -10.4 (8.5) | -12.2 (8.6) | -9.2 (10.3) | -11.1 (8.5) | -12.4 (8.9)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -10.2 (8.6) | -11.7 (8.4) | -10.1 (9.5) | -11.5 (8.1) | -12.6 (8.6)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -10.5 (8.5) | -11.8 (8.8) | -9.9 (9.6) | -12.2 (8.4) | -12.9 (8.8)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -10.6 (8.2) | -12.0 (8.7) | -10.7 (10.0) | -12.5 (7.8) | -12.8 (9.0)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -10.1 (7.1) | -12.4 (9.5) | -11.3 (9.6) | -13.2 (7.7) | -12.8 (8.7)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -10.1 (7.6) | -12.8 (9.3) | -11.4 (10.1) | -12.9 (7.9) | -12.8 (8.9)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -9.1 (9.7) | -11.5 (9.9) | -9.6 (10.7) | -11.9 (8.5) | -11.9 (8.8)

13. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) (66 Joints) at Week 12
Description: The following 66 joints subjects to assessment were examined for swollen joints and the location was confirmed. Higher SJC66 indicated greater disease activity.
  Temporomandibular joints (2), sternoclavicular joints (2), acromioclavicular joints (2), shoulder joints (2), elbow joints (2), wrist joints (2), distal interphalangeal joints (8), proximal interphalangeal joints of both hands (10), metacarpophalangeal joints (10), knee joints (2), ankle joints (2), tarsal bones (2), metatarsophalangeal joints (10), interphalangeal joint joints of toes (2), proximal interphalangeal joints of both feet (8).
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Tender Joints | -3.2 (6.0) | -6.0 (6.4) | -8.4 (5.9) | -8.3 (5.5)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -3.0, 95% CI 2-sided [-4.6 to -1.4], Standard Error of Mean 0.8 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -5.3, 95% CI 2-sided [-6.8 to -3.9], Standard Error of Mean 0.7 — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: Change From Baseline in SJC (66 Joints) Through Week 52
Description: as for outcome 13
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Swollen Joints
Groups:
- Lacebo / Peficitinib 150 mg: Participants were assigned to receive placebo to peficitinib once a day until week 12 and peficitinib 150 mg/day from week 12 to week 52.
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Lacebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Swollen Joints
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -4.5 (4.9) | -4.7 (4.2) | -2.5 (6.0) | -2.2 (4.5) | -6.3 (5.8)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -5.6 (5.6) | -7.1 (5.2) | -2.8 (5.8) | -3.4 (4.7) | -7.6 (5.2)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -6.4 (5.8) | -8.7 (6.0) | -3.3 (6.7) | -3.9 (5.6) | -8.3 (5.5)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -7.7 (6.0) | -8.7 (6.0) | -6.4 (6.3) | -6.3 (5.3) | -8.7 (5.3)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -7.6 (6.3) | -9.1 (6.2) | -6.6 (6.4) | -7.8 (6.9) | -9.2 (5.5)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 46 | 182
  Week 24 | -7.9 (6.0) | -9.7 (6.5) | -6.5 (6.2) | -8.2 (7.6) | -9.1 (5.3)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -8.2 (5.6) | -10.4 (5.7) | -6.7 (7.5) | -8.7 (7.4) | -9.7 (5.9)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -8.2 (6.3) | -10.4 (5.7) | -5.9 (8.3) | -8.2 (7.5) | -9.8 (6.1)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -8.4 (6.1) | -10.4 (6.1) | -7.6 (7.1) | -8.5 (7.7) | -9.8 (6.0)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -8.4 (5.7) | -10.4 (6.3) | -7.6 (7.0) | -9.1 (8.0) | -10.0 (6.2)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -8.8 (5.5) | -10.5 (6.2) | -8.0 (8.0) | -9.3 (8.0) | -9.9 (6.4)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -8.6 (5.8) | -10.8 (6.4) | -8.0 (7.2) | -9.1 (8.1) | -9.9 (6.0)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -8.7 (5.9) | -11.0 (6.0) | -8.2 (8.7) | -9.4 (8.0) | -10.2 (6.5)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -7.7 (7.1) | -10.0 (6.5) | -6.7 (9.7) | -8.6 (8.0) | -9.7 (6.4)

15. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP < 2.6 at Week 12
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to below description.
  DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. If the DAS28 score was less than 2.6, the participant was considered to be in DAS28 remission.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 102 | 101 | 200
Percentage of Participants | 5.0 | 24.5 | 34.7 | 45.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 6.40, 95% CI 2-sided [2.31 to 17.67] — Based on logistic regression model: DAS28-CRP score < 2.6 (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 10.13, 95% CI 2-sided [3.76 to 27.27] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP < 2.6 Through Week 52
Description: as for outcome 15
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 10.2 | 5.0 | 0.0 | 2.1 | 26.0
  Week 8: number analyzed (Participants) | 96 | 98 | 43 | 47 | 195
  Week 8 | 19.8 | 23.5 | 9.3 | 2.1 | 37.4
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 191
  Week 12 | 25.0 | 37.0 | 7.1 | 4.3 | 47.6
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 47 | 188
  Week 16 | 35.5 | 39.8 | 21.4 | 23.4 | 53.2
  Week 20: number analyzed (Participants) | 92 | 92 | 42 | 46 | 182
  Week 20 | 37.0 | 51.1 | 16.7 | 32.6 | 59.3
  Week 24: number analyzed (Participants) | 87 | 89 | 40 | 45 | 182
  Week 24 | 37.9 | 51.7 | 25.0 | 33.3 | 59.9
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 177
  Week 28 | 36.1 | 55.1 | 34.1 | 41.3 | 61.6
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 45 | 176
  Week 32 | 38.3 | 55.8 | 37.8 | 37.8 | 68.2
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 43 | 175
  Week 36 | 49.4 | 54.7 | 43.2 | 39.5 | 61.7
  Week 40: number analyzed (Participants) | 75 | 86 | 38 | 42 | 173
  Week 40 | 45.3 | 53.5 | 36.8 | 45.2 | 68.8
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | 46.7 | 57.6 | 48.6 | 41.0 | 69.6
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 43.2 | 61.9 | 51.4 | 56.4 | 70.8
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 38 | 162
  Week 52 | 43.7 | 66.7 | 45.7 | 55.3 | 67.9
  EOT: number analyzed (Participants) | 102 | 101 | 43 | 47 | 200
  EOT | 39.2 | 59.4 | 41.9 | 51.1 | 61.5

17. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR < 2.6 at Week 12
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to below description.
  DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. If the DAS28 score was less than 2.6, the participant was considered to be in DAS28 remission.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 103 | 101 | 199
Percentage of Participants | 1.0 | 11.7 | 17.8 | 31.7
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo. Difference vs. Peficitinib 100mg was not estimable; Test type: Superiority; p = 0.003, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 21.72, 95% CI 2-sided [2.83 to 166.66] — Based on logistic regression model: DAS28-ESR score < 2.6 (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)

18. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR < 2.6 Through Week 52
Description: as for outcome 17
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 2.0 | 4.0 | 0.0 | 2.1 | 14.5
  Week 8: number analyzed (Participants) | 95 | 98 | 43 | 46 | 195
  Week 8 | 8.4 | 13.3 | 0.0 | 0.0 | 27.7
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 190
  Week 12 | 11.5 | 19.6 | 2.4 | 0.0 | 33.2
  Week 16: number analyzed (Participants) | 93 | 92 | 42 | 47 | 188
  Week 16 | 18.3 | 26.1 | 11.9 | 14.9 | 35.1
  Week 20: number analyzed (Participants) | 91 | 91 | 41 | 46 | 181
  Week 20 | 22.0 | 28.6 | 14.6 | 19.6 | 38.1
  Week 24: number analyzed (Participants) | 87 | 88 | 39 | 45 | 181
  Week 24 | 23.0 | 34.1 | 15.4 | 17.8 | 41.4
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 176
  Week 28 | 27.7 | 34.8 | 26.8 | 21.7 | 39.8
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 175
  Week 32 | 22.2 | 30.2 | 19.4 | 24.4 | 43.4
  Week 36: number analyzed (Participants) | 79 | 85 | 36 | 43 | 175
  Week 36 | 25.3 | 41.2 | 25.0 | 18.6 | 40.0
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | 28.9 | 44.2 | 32.4 | 28.6 | 43.9
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 32.0 | 48.2 | 35.3 | 28.2 | 43.3
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 24.3 | 39.3 | 37.1 | 38.5 | 47.6
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 25.4 | 34.6 | 29.4 | 28.9 | 43.2
  EOT: number analyzed (Participants) | 103 | 101 | 42 | 47 | 200
  EOT | 23.3 | 28.7 | 26.2 | 27.7 | 39.5

19. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <= 3.2 at Week 12
Description: DAS28-CRP response consisted of following parameters: TJC (28 joints), SJC (28 joints), CRP, SGA, and calculated according to below description.
  DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP + 1) + 0.014 × SGA + 0.96. DAS28-CRP scores range from 0.96 to approximately 10. DAS28 score of less than or equal to 3.2 was considered to be low disease activity.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 102 | 101 | 200
Percentage of Participants | 11.0 | 40.2 | 53.5 | 68.0
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 5.80, 95% CI 2-sided [2.74 to 12.29] — Based on logistic regression model: DAS28-CRP score ≤ 3.2 (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 9.66, 95% CI 2-sided [4.57 to 20.41] — [estimate comment as in outcome 19, analysis 1]

20. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <= 3.2 Through Week 52
Description: as for outcome 19
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 18.4 | 21.0 | 4.7 | 4.3 | 47.0
  Week 8: number analyzed (Participants) | 96 | 98 | 43 | 47 | 195
  Week 8 | 32.3 | 40.8 | 11.6 | 12.8 | 59.5
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 191
  Week 12 | 41.7 | 55.4 | 14.3 | 10.6 | 70.2
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 47 | 188
  Week 16 | 52.7 | 64.5 | 33.3 | 44.7 | 73.4
  Week 20: number analyzed (Participants) | 92 | 92 | 42 | 46 | 182
  Week 20 | 55.4 | 67.4 | 45.2 | 47.8 | 75.8
  Week 24: number analyzed (Participants) | 87 | 89 | 40 | 45 | 182
  Week 24 | 50.6 | 74.2 | 35.0 | 62.2 | 77.5
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 177
  Week 28 | 55.4 | 76.4 | 41.5 | 63.0 | 81.9
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 45 | 176
  Week 32 | 58.0 | 70.9 | 51.4 | 55.6 | 83.0
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 43 | 175
  Week 36 | 63.3 | 75.6 | 56.8 | 67.4 | 83.4
  Week 40: number analyzed (Participants) | 75 | 86 | 38 | 42 | 173
  Week 40 | 62.7 | 76.7 | 57.9 | 71.4 | 85.0
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | 61.3 | 75.3 | 57.1 | 74.4 | 83.0
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 64.9 | 81.0 | 60.0 | 79.5 | 86.3
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 38 | 162
  Week 52 | 63.4 | 84.0 | 54.3 | 81.6 | 89.5
  EOT: number analyzed (Participants) | 102 | 101 | 43 | 47 | 200
  EOT | 54.9 | 77.2 | 48.8 | 76.6 | 81.5

21. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <= 3.2 at Week 12
Description: DAS28-ESR response consisted of following parameters: TJC (28 joints), SJC (28 joints), ESR, SGA , and calculated according to below description.
  DAS28 = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 × SGA. DAS28-ESR scores range from 0 to approximately 10. DAS28 score of less than or equal to 3.2 was considered to be low disease activity.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 103 | 101 | 199
Percentage of Participants | 7.0 | 19.4 | 37.6 | 49.7
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.012, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.29 to 8.12] — Based on logistic regression model: DAS28-ESR score ≤ 3.2 (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 8.19, 96% CI 2-sided [3.42 to 19.63] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <= 3.2 Through Week 52
Description: as for outcome 21
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 9.2 | 10.0 | 0.0 | 4.3 | 33.0
  Week 8: number analyzed (Participants) | 95 | 98 | 43 | 46 | 195
  Week 8 | 20.0 | 24.5 | 9.3 | 2.2 | 42.6
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 190
  Week 12 | 19.8 | 39.1 | 7.1 | 8.5 | 51.1
  Week 16: number analyzed (Participants) | 93 | 92 | 42 | 47 | 188
  Week 16 | 32.3 | 42.4 | 21.4 | 25.5 | 53.7
  Week 20: number analyzed (Participants) | 91 | 91 | 41 | 46 | 181
  Week 20 | 36.3 | 51.6 | 19.5 | 34.8 | 56.9
  Week 24: number analyzed (Participants) | 87 | 88 | 39 | 45 | 181
  Week 24 | 37.9 | 50.0 | 23.1 | 37.8 | 58.6
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 176
  Week 28 | 36.1 | 59.6 | 36.6 | 41.3 | 60.8
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 175
  Week 32 | 42.0 | 54.7 | 38.9 | 40.0 | 65.7
  Week 36: number analyzed (Participants) | 79 | 85 | 36 | 43 | 175
  Week 36 | 48.1 | 61.2 | 41.7 | 37.2 | 62.3
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | 51.3 | 59.3 | 43.2 | 47.6 | 67.1
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 48.0 | 60.0 | 50.0 | 46.2 | 64.3
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 45.9 | 61.9 | 54.3 | 53.8 | 72.6
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 45.1 | 69.1 | 41.2 | 52.6 | 62.3
  EOT: number analyzed (Participants) | 103 | 101 | 42 | 47 | 200
  EOT | 38.8 | 61.4 | 38.1 | 46.8 | 58.0

23. Secondary Outcome: Change From Baseline in CRP at Week 12
Description: Higher CRP indicates greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 101 | 101 | 200
mg/dL | 0.022 (1.498) | -1.056 (1.908) | -1.734 (1.906) | -1.207 (2.694)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS Mean = -1.112, 95% CI 2-sided [-1.546 to -0.679], Standard Error of Mean 0.220 — Based on analysis of covariance model: CRP Change = Treatment + Baseline CRP + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -1.677, 95% CI 2-sided [-2.114 to -1.241], Standard Error of Mean 0.221 — [estimate comment as in outcome 23, analysis 1]

24. Secondary Outcome: Change From Baseline in CRP Through Week 52
Description: Higher CRP indicates greater disease activity.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
mg/dL
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | -0.817 (1.566) | -1.359 (1.575) | 0.013 (1.070) | 0.073 (1.643) | -1.360 (1.511)
  Week 8: number analyzed (Participants) | 96 | 98 | 43 | 47 | 195
  Week 8 | -0.967 (1.877) | -1.664 (1.768) | 0.198 (1.662) | -0.076 (0.930) | -1.337 (1.822)
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 192
  Week 12 | -1.045 (1.827) | -1.810 (1.908) | 0.026 (1.852) | -0.142 (1.076) | -1.205 (2.735)
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 47 | 188
  Week 16 | -1.083 (2.062) | -1.849 (2.099) | -0.802 (2.127) | -1.180 (1.109) | -1.383 (1.639)
  Week 20: number analyzed (Participants) | 92 | 92 | 42 | 46 | 182
  Week 20 | -0.964 (2.551) | -1.819 (2.156) | -0.581 (2.471) | -1.294 (1.152) | -1.525 (1.643)
  Week 24: number analyzed (Participants) | 87 | 89 | 40 | 45 | 182
  Week 24 | -1.225 (2.168) | -1.824 (2.200) | -0.434 (2.251) | -1.318 (1.486) | -1.473 (1.847)
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 177
  Week 28 | -1.323 (1.976) | -1.904 (2.197) | -1.013 (2.247) | -1.266 (1.635) | -1.611 (2.000)
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 45 | 176
  Week 32 | -1.200 (1.973) | -1.979 (2.223) | -1.239 (2.227) | -0.975 (3.345) | -1.593 (1.886)
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 43 | 175
  Week 36 | -1.310 (1.874) | -2.043 (2.202) | -1.084 (2.460) | -1.192 (1.453) | -1.467 (2.233)
  Week 40: number analyzed (Participants) | 75 | 86 | 38 | 42 | 173
  Week 40 | -1.199 (2.011) | -2.019 (2.240) | -1.325 (2.566) | -1.232 (1.609) | -1.594 (2.146)
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | -1.202 (1.961) | -1.978 (2.221) | -1.292 (2.366) | -1.225 (1.729) | -1.627 (1.810)
  Week 48: number analyzed (Participants) | 75 | 84 | 35 | 39 | 168
  Week 48 | -0.964 (2.074) | -1.833 (2.882) | -1.610 (2.103) | -1.407 (1.747) | -1.611 (1.858)
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 38 | 162
  Week 52 | -1.138 (2.056) | -2.068 (2.228) | -1.566 (2.034) | -1.534 (1.589) | -1.595 (1.873)
  EOT: number analyzed (Participants) | 101 | 101 | 43 | 47 | 200
  EOT | -0.949 (2.368) | -1.832 (2.221) | -0.797 (2.879) | -0.987 (3.366) | -1.326 (2.724)

25. Secondary Outcome: Change From Baseline in ESR at Week 12
Description: Higher ESR indicates greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 199
mm/hour | -1.96 (17.82) | -12.96 (21.51) | -23.92 (21.26) | -20.92 (21.66)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -10.90, 95% CI 2-sided [-15.95 to -5.84], Standard Error of Mean 2.56 — Based on analysis of covariance model: ESR Change = Treatment + Baseline ESR + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -21.14, 95% CI 2-sided [-26.01 to -16.27], Standard Error of Mean 2.47 — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Change From Baseline in ESR Through Week 52
Description: Higher ESR indicates greater disease activity.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
mm/hour
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 46 | 199
  Week 4 | -9.98 (15.44) | -14.99 (15.90) | -0.63 (11.77) | -3.87 (12.99) | -19.20 (17.51)
  Week 8: number analyzed (Participants) | 96 | 98 | 43 | 46 | 194
  Week 8 | -15.27 (19.29) | -21.59 (19.81) | -0.95 (12.47) | -2.07 (14.31) | -20.88 (19.43)
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 46 | 191
  Week 12 | -13.49 (21.25) | -25.26 (21.22) | -2.62 (18.31) | -4.43 (17.07) | -21.74 (20.67)
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 46 | 188
  Week 16 | -15.34 (20.98) | -28.32 (21.66) | -11.76 (19.87) | -16.89 (17.70) | -22.05 (19.53)
  Week 20: number analyzed (Participants) | 91 | 92 | 42 | 45 | 182
  Week 20 | -16.77 (21.88) | -27.34 (21.95) | -12.69 (23.03) | -20.62 (17.65) | -21.91 (20.59)
  Week 24: number analyzed (Participants) | 87 | 89 | 40 | 45 | 182
  Week 24 | -17.61 (22.60) | -27.02 (26.00) | -13.18 (21.90) | -20.04 (18.45) | -22.20 (23.87)
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 45 | 177
  Week 28 | -16.47 (21.90) | -27.21 (23.97) | -16.29 (17.77) | -18.02 (24.26) | -23.52 (22.35)
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 44 | 176
  Week 32 | -16.35 (23.09) | -27.02 (23.81) | -19.54 (21.98) | -19.93 (25.80) | -24.75 (21.27)
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 42 | 175
  Week 36 | -18.67 (23.77) | -29.50 (25.26) | -19.65 (22.64) | -21.99 (21.52) | -24.66 (22.32)
  Week 40: number analyzed (Participants) | 76 | 86 | 38 | 41 | 173
  Week 40 | -17.74 (25.65) | -29.79 (24.00) | -19.45 (23.06) | -21.71 (25.48) | -25.87 (24.84)
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | -17.77 (25.35) | -29.07 (24.47) | -21.43 (24.12) | -22.31 (23.12) | -25.73 (21.09)
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 38 | 168
  Week 48 | -15.43 (25.70) | -28.70 (24.69) | -23.40 (23.87) | -25.66 (22.30) | -25.98 (22.00)
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 37 | 162
  Week 52 | -16.77 (26.05) | -28.59 (24.97) | -21.03 (19.81) | -23.24 (24.28) | -24.23 (21.70)
  EOT: number analyzed (Participants) | 102 | 101 | 43 | 46 | 199
  EOT | -14.94 (27.20) | -26.15 (25.02) | -15.37 (24.27) | -18.61 (27.67) | -20.75 (26.25)

27. Secondary Outcome: Percentage of Participants With a European League Against Rheumatism (EULAR) Good Response Using DAS28-CRP at Week 12
Description: Good response was defined as DAS28 after treatment ≤ 3.2 and improvement from baseline > 1.2.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 101 | 101 | 200
Percentage of Participants | 9.1 | 38.6 | 51.5 | 65.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 6.64, 95% CI 2-sided [2.98 to 14.83] — Based on logistic regression model: Good Response (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 10.86, 95% CI 2-sided [4.91 to 24.03] — [estimate comment as in outcome 27, analysis 1]

28. Secondary Outcome: Percentage of Participants With a EULAR Good Response Using DAS28-CRP Through Week 52
Description: Good response was defined as DAS28 after treatment ≤ 3.2 and improvement from baseline > 1.2.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | 17.3 | 16.0 | 4.8 | 2.1 | 44.5
  Week 8: number analyzed (Participants) | 96 | 98 | 42 | 47 | 195
  Week 8 | 28.1 | 39.8 | 11.9 | 6.4 | 56.4
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | 39.6 | 53.3 | 12.2 | 8.5 | 67.5
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | 48.4 | 60.2 | 34.1 | 40.4 | 72.9
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | 51.1 | 65.2 | 46.3 | 43.5 | 75.8
  Week 24: number analyzed (Participants) | 87 | 89 | 39 | 45 | 182
  Week 24 | 47.1 | 71.9 | 33.3 | 57.8 | 76.4
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | 50.6 | 74.2 | 40.0 | 58.7 | 80.8
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | 54.3 | 68.6 | 50.0 | 46.7 | 83.0
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | 59.5 | 74.4 | 55.6 | 62.8 | 83.4
  Week 40: number analyzed (Participants) | 75 | 86 | 37 | 42 | 173
  Week 40 | 58.7 | 75.6 | 54.1 | 66.7 | 84.4
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 58.7 | 74.1 | 55.9 | 71.8 | 82.5
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | 60.8 | 79.8 | 55.9 | 79.5 | 85.1
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 59.2 | 81.5 | 52.9 | 78.9 | 88.3
  EOT: number analyzed (Participants) | 101 | 101 | 42 | 47 | 200
  EOT | 52.5 | 75.2 | 47.6 | 72.3 | 80.0

29. Secondary Outcome: Percentage of Participants With a Good or Moderate EULAR Response Using DAS28-CRP at Week 12
Description: Good and moderate response was defined as DAS28 after treatment ≤ 5.1 and improvement from baseline > 0.6, or DAS28 after treatment > 5.1 and improvement from baseline > 1.2.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 101 | 101 | 200
Percentage of Participants | 41.4 | 75.2 | 92.1 | 92.5
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 4.37, 95% CI 2-sided [2.38 to 8.04] — Based on logistic regression model: Good or Moderate Response (responder, non-responder) = Treatment + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 16.78, 95% CI 2-sided [7.31 to 38.51] — [estimate comment as in outcome 29, analysis 1]

30. Secondary Outcome: Percentage of Participants With a Good or Moderate EULAR Response Using DAS28-CRP Through Week 52
Description: as for outcome 29
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | 63.3 | 72.0 | 31.0 | 40.4 | 87.5
  Week 8: number analyzed (Participants) | 96 | 98 | 42 | 47 | 195
  Week 8 | 76.0 | 86.7 | 47.6 | 40.4 | 92.3
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | 77.1 | 94.6 | 41.5 | 48.9 | 94.2
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | 81.7 | 92.5 | 73.2 | 85.1 | 96.8
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | 79.3 | 96.7 | 78.0 | 91.3 | 95.6
  Week 24: number analyzed (Participants) | 87 | 89 | 39 | 45 | 182
  Week 24 | 85.1 | 96.6 | 71.8 | 91.1 | 97.3
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | 89.2 | 95.5 | 80.0 | 87.0 | 99.4
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | 91.4 | 96.5 | 83.3 | 82.2 | 98.3
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | 87.3 | 96.5 | 86.1 | 86.0 | 97.7
  Week 40: number analyzed (Participants) | 75 | 86 | 37 | 42 | 173
  Week 40 | 89.3 | 96.5 | 86.5 | 85.7 | 100.0
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | 93.3 | 94.1 | 88.2 | 87.2 | 99.4
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | 90.5 | 97.6 | 94.1 | 89.7 | 98.2
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | 91.5 | 98.8 | 94.1 | 92.1 | 98.8
  EOT: number analyzed (Participants) | 101 | 101 | 42 | 47 | 200
  EOT | 78.2 | 93.1 | 83.3 | 85.1 | 95.5

31. Secondary Outcome: Percentage of Participants With a Good EULAR Response Using DAS28-ESR at Week 12
Description: Good response was defined as DAS28 after treatment ≤ 3.2 and improvement from baseline > 1.2.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 98 | 102 | 101 | 198
Percentage of Participants | 5.1 | 18.6 | 36.6 | 49.0
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.006, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 4.29, 95% CI 2-sided [1.52 to 12.08] — [estimate comment as in outcome 27, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio, log = 11.01, 95% CI 2-sided [4.07 to 29.74] — [estimate comment as in outcome 27, analysis 1]

32. Secondary Outcome: Percentage of Participants With a Good EULAR Response Using DAS28-ESR Through Week 52
Description: Good response was defined as DAS28 after treatment ≤ 3.2 and improvement from baseline > 1.2.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 46 | 199
  Week 4 | 8.2 | 10.0 | 0.0 | 2.2 | 31.7
  Week 8: number analyzed (Participants) | 95 | 98 | 42 | 45 | 194
  Week 8 | 16.8 | 24.5 | 9.5 | 0.0 | 41.2
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 46 | 190
  Week 12 | 18.8 | 38.0 | 4.9 | 6.5 | 50.0
  Week 16: number analyzed (Participants) | 93 | 92 | 41 | 46 | 188
  Week 16 | 31.2 | 40.2 | 22.0 | 21.7 | 52.7
  Week 20: number analyzed (Participants) | 91 | 91 | 40 | 45 | 181
  Week 20 | 34.1 | 51.6 | 20.0 | 31.1 | 56.4
  Week 24: number analyzed (Participants) | 87 | 88 | 38 | 44 | 181
  Week 24 | 35.6 | 50.0 | 21.1 | 34.1 | 56.4
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 45 | 176
  Week 28 | 32.5 | 59.6 | 35.0 | 37.8 | 59.7
  Week 32: number analyzed (Participants) | 81 | 86 | 35 | 44 | 175
  Week 32 | 39.5 | 54.7 | 37.1 | 36.4 | 63.4
  Week 36: number analyzed (Participants) | 79 | 85 | 35 | 42 | 175
  Week 36 | 44.3 | 60.0 | 40.0 | 33.3 | 62.3
  Week 40: number analyzed (Participants) | 76 | 86 | 36 | 41 | 173
  Week 40 | 47.4 | 59.3 | 41.7 | 43.9 | 67.1
  Week 44: number analyzed (Participants) | 75 | 85 | 33 | 39 | 171
  Week 44 | 45.3 | 60.0 | 48.5 | 43.6 | 63.7
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 38 | 168
  Week 48 | 41.9 | 61.9 | 52.9 | 52.6 | 72.6
  Week 52: number analyzed (Participants) | 71 | 81 | 33 | 37 | 162
  Week 52 | 43.7 | 69.1 | 39.4 | 48.6 | 61.7
  EOT: number analyzed (Participants) | 102 | 101 | 41 | 46 | 199
  EOT | 38.2 | 61.4 | 36.6 | 43.5 | 57.3

33. Secondary Outcome: Percentage of Participants With a Good or Moderate EULAR Response Using DAS28-ESR at Week 12
Description: as for outcome 29
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 98 | 102 | 101 | 198
Percentage of Participants | 37.8 | 69.6 | 88.1 | 90.9
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 3.82, 95% CI [2.11 to 6.93] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Wald's chi-squared test — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = 13.65, 95% CI 2-sided [6.39 to 29.17] — [estimate comment as in outcome 29, analysis 1]

34. Secondary Outcome: Percentage of Participants With a Good or Moderate EULAR Response Using DAS28-ESR Through Week 52
Description: as for outcome 29
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 46 | 199
  Week 4 | 56.1 | 65.0 | 31.0 | 23.9 | 81.9
  Week 8: number analyzed (Participants) | 95 | 98 | 42 | 45 | 194
  Week 8 | 66.3 | 84.7 | 45.2 | 33.3 | 92.8
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 46 | 190
  Week 12 | 70.8 | 90.2 | 39.0 | 43.5 | 92.6
  Week 16: number analyzed (Participants) | 93 | 92 | 41 | 46 | 188
  Week 16 | 76.3 | 88.0 | 73.2 | 76.1 | 94.7
  Week 20: number analyzed (Participants) | 91 | 91 | 40 | 45 | 181
  Week 20 | 79.1 | 96.7 | 72.5 | 86.7 | 93.9
  Week 24: number analyzed (Participants) | 87 | 88 | 38 | 44 | 181
  Week 24 | 82.8 | 95.5 | 73.7 | 90.9 | 96.1
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 45 | 176
  Week 28 | 84.3 | 92.1 | 77.5 | 88.9 | 97.7
  Week 32: number analyzed (Participants) | 81 | 86 | 35 | 44 | 175
  Week 32 | 90.1 | 94.2 | 77.1 | 86.4 | 97.1
  Week 36: number analyzed (Participants) | 79 | 85 | 35 | 42 | 175
  Week 36 | 83.5 | 95.3 | 85.7 | 83.3 | 96.6
  Week 40: number analyzed (Participants) | 76 | 86 | 36 | 41 | 173
  Week 40 | 89.5 | 95.3 | 83.3 | 85.4 | 98.3
  Week 44: number analyzed (Participants) | 75 | 85 | 33 | 39 | 171
  Week 44 | 90.7 | 92.9 | 84.8 | 87.2 | 98.2
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 38 | 168
  Week 48 | 86.5 | 95.2 | 88.2 | 89.5 | 98.2
  Week 52: number analyzed (Participants) | 71 | 81 | 33 | 37 | 162
  Week 52 | 84.5 | 97.5 | 84.8 | 89.2 | 98.1
  EOT: number analyzed (Participants) | 102 | 101 | 41 | 46 | 199
  EOT | 74.5 | 94.1 | 75.6 | 82.6 | 93.5

35. Secondary Outcome: Percentage of Participants Achieving ACR / EULAR Remission at Week 12
Description: ACR/EULAR Remission was defined as TJC (68 joints) ≤ 1, SJC (66 joints) ≤ 1, CRP ≤ 1 mg/dL, and subject's global assessment of arthritis ≤ 1 cm (on a visual analog scale (VAS) of 0 - 100 mm).
  Statistical analysis of treatment difference vs placebo was not estimable for either peficitinib 100 mg or peficitinib 150 mg reporting groups.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 102 | 101 | 200
Percentage of Participants | 2.0 | 5.9 | 5.9 | 13.5

36. Secondary Outcome: Percentage of Participants Achieving ACR / EULAR Remission Through Week 52
Description: ACR/EULAR Remission was defined as TJC (68 joints) ≤ 1, SJC (66 joints) ≤ 1, CRP ≤ 1 mg/dL, and subject's global assessment of arthritis ≤ 1 cm (on a VAS of 0 - 100 mm).
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 1.0 | 0.0 | 0.0 | 0.0 | 7.0
  Week 8: number analyzed (Participants) | 96 | 98 | 43 | 47 | 195
  Week 8 | 2.1 | 1.0 | 2.3 | 0.0 | 11.8
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 191
  Week 12 | 6.3 | 6.5 | 0.0 | 4.3 | 14.1
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 47 | 188
  Week 16 | 11.8 | 8.6 | 4.8 | 2.1 | 18.6
  Week 20: number analyzed (Participants) | 92 | 92 | 42 | 46 | 182
  Week 20 | 12.0 | 13.0 | 4.8 | 6.5 | 20.9
  Week 24: number analyzed (Participants) | 87 | 89 | 40 | 45 | 182
  Week 24 | 13.8 | 10.1 | 5.0 | 8.9 | 28.0
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 177
  Week 28 | 12.0 | 18.0 | 9.8 | 10.9 | 24.3
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 45 | 176
  Week 32 | 13.6 | 20.9 | 10.8 | 11.1 | 25.0
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 43 | 175
  Week 36 | 16.5 | 18.6 | 8.1 | 7.0 | 22.3
  Week 40: number analyzed (Participants) | 75 | 86 | 38 | 42 | 173
  Week 40 | 16.0 | 19.8 | 7.9 | 14.3 | 24.3
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | 16.0 | 24.7 | 20.0 | 7.7 | 25.1
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 17.6 | 25.0 | 25.7 | 15.4 | 27.4
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 38 | 162
  Week 52 | 18.3 | 18.5 | 22.9 | 10.5 | 30.2
  EOT: number analyzed (Participants) | 102 | 101 | 43 | 47 | 200
  EOT | 14.7 | 15.8 | 20.9 | 8.5 | 25.0

37. Secondary Outcome: Percentage of Participants Achieving Simplified Disease Activity Index (SDAI) Remission at Week 12
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to below description.
  SDAI = TJC + SJC + SGA + PGA + CRP. SDAI Remission was defined as SDAI score ≤ 3.3.
  Statistical analysis of treatment difference vs placebo was not estimable for either peficitinib 100 mg or peficitinib 150 mg reporting groups.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 102 | 101 | 200
Percentage of Participants | 0.0 | 8.8 | 8.9 | 18.5

38. Secondary Outcome: Percentage of Participants Achieving SDAI Remission Through Week 52
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to below description.
  SDAI = TJC + SJC + SGA + PGA + CRP. SDAI Remission was defined as SDAI score ≤ 3.3.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 1.0 | 1.0 | 0.0 | 0.0 | 10.0
  Week 8: number analyzed (Participants) | 96 | 98 | 43 | 47 | 195
  Week 8 | 4.2 | 6.1 | 0.0 | 0.0 | 16.9
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 191
  Week 12 | 9.4 | 9.8 | 0.0 | 0.0 | 19.4
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 47 | 188
  Week 16 | 12.9 | 15.1 | 2.4 | 8.5 | 23.9
  Week 20: number analyzed (Participants) | 92 | 92 | 42 | 46 | 182
  Week 20 | 17.4 | 18.5 | 4.8 | 15.2 | 29.7
  Week 24: number analyzed (Participants) | 87 | 89 | 40 | 45 | 182
  Week 24 | 18.4 | 18.0 | 10.0 | 17.8 | 34.1
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 177
  Week 28 | 19.3 | 29.2 | 17.1 | 17.4 | 33.9
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 45 | 176
  Week 32 | 16.0 | 27.9 | 13.5 | 13.3 | 35.2
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 43 | 175
  Week 36 | 21.5 | 27.9 | 18.9 | 4.7 | 30.9
  Week 40: number analyzed (Participants) | 75 | 86 | 38 | 42 | 173
  Week 40 | 24.0 | 36.0 | 10.5 | 19.0 | 33.5
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | 22.7 | 38.8 | 20.0 | 15.4 | 34.5
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 18.9 | 38.1 | 28.6 | 25.6 | 39.3
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 38 | 162
  Week 52 | 21.1 | 29.6 | 20.0 | 21.1 | 39.5
  EOT: number analyzed (Participants) | 102 | 101 | 43 | 47 | 200
  EOT | 17.6 | 25.7 | 18.6 | 17.0 | 33.5

39. Secondary Outcome: Change From Baseline in SDAI Score at Week 12
Description: SDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, CRP (mg/dL), and calculated according to below description.
  SDAI = TJC + SJC + SGA + PGA + CRP. The SDAI score ranges from 0 to approximately 86. Higher SDAI indicates greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 101 | 101 | 200
Units on a Scale | -7.22 (14.11) | -16.08 (14.37) | -20.93 (11.32) | -21.94 (11.21)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS Mean = -9.94, 95% CI 2-sided [-13.66 to -6.22], Standard Error of Mean 1.89 — Based on analysis of covariance model: SDAI Change = Treatment + Baseline SDAI + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; Odds Ratio (OR) = -14.43, 95% CI 2-sided [-17.71 to -11.15], Standard Error of Mean 1.66 — [estimate comment as in outcome 39, analysis 1]

40. Secondary Outcome: Change From Baseline in SDAI Score Through Week 52
Description: as for outcome 39
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -11.83 (9.97) | -12.78 (9.06) | -5.57 (9.50) | -7.21 (9.35) | -17.09 (10.83)
  Week 8: number analyzed (Participants) | 96 | 98 | 42 | 47 | 195
  Week 8 | -14.71 (12.53) | -18.66 (9.73) | -7.07 (12.26) | -8.43 (11.37) | -20.64 (10.09)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -16.59 (13.47) | -21.62 (11.48) | -7.48 (14.80) | -10.18 (11.82) | -22.54 (10.79)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -19.25 (13.76) | -21.90 (12.19) | -15.20 (14.25) | -18.90 (12.08) | -23.46 (10.37)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -19.47 (14.16) | -23.37 (11.94) | -15.67 (15.41) | -20.61 (12.44) | -24.44 (10.15)
  Week 24: number analyzed (Participants) | 87 | 89 | 39 | 45 | 182
  Week 24 | -20.14 (13.96) | -24.40 (12.00) | -16.13 (14.40) | -22.25 (13.22) | -24.78 (10.14)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -20.29 (12.71) | -25.29 (12.32) | -17.75 (15.21) | -22.74 (13.00) | -25.70 (10.51)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -21.72 (12.82) | -25.28 (12.07) | -17.71 (15.34) | -21.14 (14.69) | -25.84 (10.79)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -21.34 (12.65) | -25.62 (11.95) | -20.57 (14.03) | -22.02 (13.54) | -25.77 (11.33)
  Week 40: number analyzed (Participants) | 75 | 86 | 37 | 42 | 173
  Week 40 | -21.55 (13.04) | -25.78 (12.54) | -20.34 (14.90) | -23.09 (14.63) | -26.46 (11.11)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -21.54 (12.22) | -25.82 (12.92) | -22.65 (13.74) | -23.23 (14.31) | -26.17 (11.06)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -21.11 (12.13) | -26.33 (12.58) | -23.21 (13.47) | -24.61 (13.35) | -26.57 (11.02)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -21.19 (12.83) | -26.99 (12.52) | -23.04 (13.57) | -25.20 (13.91) | -26.77 (11.57)
  EOT: number analyzed (Participants) | 101 | 101 | 42 | 47 | 200
  EOT | -18.92 (15.76) | -24.95 (12.77) | -18.76 (16.83) | -22.38 (15.91) | -24.85 (12.19)

41. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Score <= 2.8 at Week 12
Description: CDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, and calculated according to below description.
  CDAI = TJC + SJC + SGA + PGA. CDAI. Remission was defined as CDAI score ≤ 2.8. Statistical analysis of treatment difference vs placebo was not estimable for either peficitinib 100 mg or peficitinib 150 mg reporting groups.
Time Frame: Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 100 | 103 | 101 | 200
Percentage of Participants | 0.0 | 8.7 | 9.9 | 19.0

42. Secondary Outcome: Percentage of Participants Achieving CDAI Score <= 2.8 Through Week 52
Description: CDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, and calculated according to below description.
  CDAI = TJC + SJC + SGA + PGA. CDAI. Remission was defined as CDAI score ≤ 2.8.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Percentage of Participants
  Week 4: number analyzed (Participants) | 98 | 100 | 43 | 47 | 200
  Week 4 | 1.0 | 2.0 | 0.0 | 0.0 | 9.0
  Week 8: number analyzed (Participants) | 96 | 99 | 43 | 47 | 195
  Week 8 | 4.2 | 6.1 | 0.0 | 0.0 | 14.4
  Week 12: number analyzed (Participants) | 96 | 92 | 42 | 47 | 191
  Week 12 | 9.4 | 10.9 | 0.0 | 0.0 | 19.9
  Week 16: number analyzed (Participants) | 93 | 93 | 42 | 47 | 188
  Week 16 | 14.0 | 16.1 | 2.4 | 6.4 | 23.9
  Week 20: number analyzed (Participants) | 92 | 92 | 42 | 46 | 182
  Week 20 | 18.5 | 17.4 | 2.4 | 10.9 | 28.0
  Week 24: number analyzed (Participants) | 87 | 90 | 40 | 45 | 182
  Week 24 | 16.1 | 15.6 | 7.5 | 15.6 | 31.9
  Week 28: number analyzed (Participants) | 83 | 89 | 41 | 46 | 177
  Week 28 | 20.5 | 27.0 | 14.6 | 17.4 | 31.6
  Week 32: number analyzed (Participants) | 81 | 86 | 37 | 45 | 176
  Week 32 | 17.3 | 27.9 | 16.2 | 13.3 | 32.4
  Week 36: number analyzed (Participants) | 79 | 86 | 37 | 43 | 175
  Week 36 | 19.0 | 26.7 | 18.9 | 7.0 | 30.3
  Week 40: number analyzed (Participants) | 76 | 86 | 38 | 42 | 173
  Week 40 | 22.4 | 29.1 | 13.2 | 21.4 | 31.8
  Week 44: number analyzed (Participants) | 75 | 85 | 35 | 39 | 171
  Week 44 | 21.3 | 36.5 | 25.7 | 15.4 | 33.3
  Week 48: number analyzed (Participants) | 74 | 84 | 35 | 39 | 168
  Week 48 | 23.0 | 34.5 | 28.6 | 23.1 | 36.3
  Week 52: number analyzed (Participants) | 71 | 81 | 35 | 38 | 162
  Week 52 | 21.1 | 27.2 | 22.9 | 18.4 | 38.3
  EOT: number analyzed (Participants) | 103 | 101 | 43 | 47 | 200
  EOT | 18.4 | 23.8 | 20.9 | 17.0 | 32.5

43. Secondary Outcome: Change From Baseline in CDAI Score at Week 12
Description: CDAI score consisted of following parameters: TJC (28 joints), SJC (28 joints), SGA, PGA, and calculated according to below description.
  CDAI = TJC + SJC + SGA + PGA. The CDAI score ranges from 0 to approximately 76. Higher CDAI indicates greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | -7.25 (13.42) | -14.91 (13.46) | -19.20 (11.04) | -20.74 (10.64)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -8.69, 95% CI 2-sided [-12.19 to -5.20], Standard Error of Mean 1.77 — Based on ANCOVA Model: CDAI Change = Treatment + Baseline CDAI + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -12.83, 95% CI 2-sided [-15.96 to -9.71], Standard Error of Mean 1.58 — [estimate comment as in outcome 43, analysis 1]

44. Secondary Outcome: Change From Baseline in CDAI Score Through Week 52
Description: as for outcome 43
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -11.01 (9.47) | -11.42 (8.99) | -5.61 (9.16) | -7.28 (8.76) | -15.73 (10.51)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -13.74 (11.77) | -17.06 (9.58) | -7.29 (11.46) | -8.35 (11.10) | -19.31 (9.69)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -15.55 (12.71) | -19.81 (11.21) | -7.52 (13.88) | -10.04 (11.47) | -21.21 (10.39)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -18.17 (12.81) | -20.06 (11.91) | -14.40 (13.13) | -17.72 (11.75) | -22.08 (10.12)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -18.51 (13.13) | -21.55 (11.42) | -15.08 (14.22) | -19.31 (12.30) | -22.92 (10.04)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | -18.92 (12.65) | -22.28 (11.75) | -15.71 (13.08) | -20.93 (12.88) | -23.30 (9.93)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -18.97 (12.06) | -23.38 (11.76) | -16.74 (14.06) | -21.48 (12.70) | -24.09 (10.26)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -20.52 (12.07) | -23.30 (11.53) | -16.46 (14.45) | -20.17 (13.87) | -24.25 (10.38)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -20.03 (12.22) | -23.58 (11.41) | -19.48 (12.86) | -20.83 (13.10) | -24.30 (10.86)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -20.41 (12.12) | -23.76 (12.03) | -19.00 (13.77) | -21.86 (14.11) | -24.87 (10.76)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -20.34 (11.43) | -23.84 (12.25) | -21.34 (12.56) | -22.00 (13.79) | -24.54 (10.81)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -20.11 (11.47) | -24.50 (11.77) | -21.58 (12.56) | -23.20 (13.03) | -24.96 (10.70)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -20.05 (11.94) | -24.93 (11.90) | -21.44 (12.72) | -23.67 (13.42) | -25.17 (11.14)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -17.82 (14.69) | -23.12 (12.04) | -17.96 (15.14) | -21.39 (14.85) | -23.52 (11.45)

45. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis (PGA) at Week 12
Description: The investigator assessed the participants' disease activity on a VAS of 0-100 mm on the physician assessment table. Higher PGA (100 mm VAS) scores indicate greater activity impairment.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | -13.94 (24.85) | -27.69 (25.39) | -34.65 (21.19) | -37.40 (20.69)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -15.20, 95% CI 2-sided [-21.40 to -9.00], Standard Error of Mean 3.14 — Based on analysis of covariance model: PGA (100 mm VAS) Change = Treatment + Baseline PGA (100 mm VAS) + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -23.14, 95% CI 2-sided [-28.78 to -17.51], Standard Error of Mean 2.86 — [estimate comment as in outcome 45, analysis 1]

46. Secondary Outcome: Change From Baseline in PGA Through Week 52
Description: as for outcome 45
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
units on a scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -18.71 (17.32) | -19.49 (18.14) | -8.77 (17.97) | -12.37 (16.60) | -27.48 (20.10)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -25.92 (23.49) | -30.55 (21.05) | -11.70 (20.42) | -16.04 (22.64) | -33.80 (19.61)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -28.91 (25.08) | -35.53 (21.28) | -14.85 (24.59) | -18.99 (23.44) | -37.99 (20.16)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -34.84 (23.77) | -34.68 (22.76) | -26.10 (22.44) | -31.35 (20.54) | -39.20 (20.77)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -34.83 (24.45) | -38.65 (21.19) | -28.43 (22.91) | -33.80 (21.18) | -41.10 (20.77)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | -36.67 (23.23) | -38.50 (23.05) | -30.62 (21.72) | -37.43 (21.86) | -41.18 (20.68)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -37.17 (22.57) | -39.29 (21.74) | -31.69 (24.41) | -37.90 (22.50) | -41.51 (20.87)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -39.14 (22.04) | -40.49 (21.08) | -30.22 (21.37) | -37.27 (23.10) | -41.95 (20.76)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -38.29 (23.55) | -40.76 (21.04) | -35.44 (22.26) | -38.90 (21.79) | -41.27 (21.41)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -39.95 (23.16) | -41.88 (21.29) | -36.31 (23.59) | -38.83 (22.58) | -42.93 (20.16)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -38.53 (22.64) | -42.16 (21.19) | -38.01 (23.72) | -37.74 (23.46) | -42.65 (20.13)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -38.29 (22.29) | -43.41 (20.74) | -39.09 (20.99) | -41.99 (22.00) | -43.71 (20.63)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -37.85 (23.45) | -44.02 (22.47) | -39.43 (21.85) | -43.24 (24.17) | -44.11 (20.69)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -34.09 (25.92) | -40.56 (22.93) | -33.01 (25.17) | -39.28 (24.37) | -41.07 (22.71)

47. Secondary Outcome: Change From Baseline in Subject's SGA at Week 12
Description: The participant assessed his/her own disease activity on a VAS of 0-100 mm on the questionnaire form. Higher SGA (100 mm VAS) scores indicate greater activity impairment.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | -7.87 (25.15) | -23.74 (32.14) | -31.59 (27.41) | -32.43 (27.39)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -16.88, 95% CI 2-sided [-23.81 to -9.95], Standard Error of Mean 3.51 — Based on analysis of covariance model: SGA (100 mm VAS) Change = Treatment + Baseline SGA (100 mm VAS) + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -23.56, 95% CI 2-sided [-29.83 to -17.28], Standard Error of Mean 3.18 — [estimate comment as in outcome 47, analysis 1]

48. Secondary Outcome: Change From Baseline in SGA Through Week 52
Description: as for outcome 47
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
units on a scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -14.66 (24.11) | -18.30 (24.25) | -1.83 (18.03) | -6.59 (21.35) | -24.38 (25.81)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -21.29 (30.24) | -29.55 (26.34) | -5.71 (22.02) | -8.78 (21.39) | -29.31 (26.07)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -25.09 (31.56) | -32.75 (27.51) | -6.93 (22.74) | -8.85 (27.24) | -33.14 (27.23)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -29.98 (30.36) | -34.37 (28.43) | -21.29 (24.56) | -21.98 (25.10) | -34.88 (25.91)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -29.82 (32.87) | -36.21 (26.97) | -17.76 (26.75) | -24.53 (24.24) | -36.10 (26.28)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | -30.09 (31.93) | -37.51 (29.32) | -25.96 (25.72) | -25.42 (26.02) | -37.12 (26.33)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -31.19 (33.76) | -37.91 (27.72) | -25.66 (27.71) | -26.01 (26.63) | -37.75 (26.52)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -34.49 (30.49) | -38.71 (28.92) | -27.97 (28.37) | -26.17 (28.46) | -38.02 (27.74)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -32.11 (30.55) | -39.08 (26.81) | -31.56 (25.36) | -26.64 (26.00) | -37.54 (27.65)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -34.66 (32.19) | -40.85 (28.00) | -30.76 (27.65) | -28.80 (28.13) | -38.42 (26.72)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -34.87 (32.36) | -39.51 (29.51) | -36.01 (27.49) | -28.19 (26.52) | -39.01 (26.58)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -35.53 (32.53) | -41.60 (27.74) | -34.09 (26.60) | -31.05 (27.81) | -39.47 (26.06)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -35.61 (33.45) | -41.54 (28.60) | -32.06 (28.15) | -32.91 (27.33) | -40.36 (27.01)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -28.52 (35.62) | -38.84 (29.05) | -26.80 (30.15) | -28.71 (27.54) | -37.09 (27.62)

49. Secondary Outcome: Change From Baseline in Subject's Assessment of Pain at Week 12
Description: The participant assessed his/her own pain severity on a VAS from 0-100 mm on the questionnaire form. Higher SGA of pain (100 mm VAS) scores indicate greater activity pain.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | -6.64 (24.61) | -23.78 (30.75) | -30.65 (27.91) | -30.82 (27.68)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -17.58, 95% CI 2-sided [-24.36 to -10.81], Standard Error of Mean 3.44 — Based on analysis of covariance model: SGA of pain (100 mm VAS) Change = Treatment + Baseline SGA of pain (100 mm VAS) + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -23.90, 95% CI 2-sided [-30.24 to -17.57], Standard Error of Mean 3.21 — [estimate comment as in outcome 49, analysis 1]

50. Secondary Outcome: Change From Baseline in Subject's Assessment of Pain Through Week 52
Description: as for outcome 49
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -14.80 (29.58) | -18.36 (24.49) | -2.00 (18.75) | -8.23 (25.32) | -22.24 (25.57)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -22.45 (31.06) | -29.58 (26.18) | -4.11 (21.26) | -9.17 (22.75) | -27.43 (26.90)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -25.02 (30.64) | -31.83 (28.13) | -5.40 (24.28) | -9.15 (25.80) | -31.37 (27.66)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -28.58 (31.83) | -34.41 (27.22) | -20.93 (25.76) | -21.20 (23.95) | -32.48 (26.22)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -29.68 (32.42) | -35.83 (28.40) | -16.21 (28.27) | -24.63 (26.52) | -34.76 (26.53)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | -29.78 (32.23) | -37.78 (28.87) | -22.64 (26.09) | -26.51 (25.46) | -35.45 (27.27)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -31.66 (31.61) | -36.48 (29.18) | -22.63 (28.92) | -24.93 (26.19) | -36.23 (27.15)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -34.15 (30.84) | -37.65 (28.66) | -25.53 (27.07) | -27.09 (26.20) | -37.20 (27.18)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -32.44 (30.76) | -38.48 (27.27) | -28.38 (25.68) | -26.79 (25.38) | -36.31 (26.59)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -35.06 (31.74) | -40.67 (27.68) | -26.65 (28.10) | -29.48 (26.77) | -36.45 (26.58)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -34.59 (30.82) | -38.76 (29.25) | -32.32 (27.16) | -28.55 (25.32) | -36.24 (25.37)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -34.87 (31.77) | -40.27 (28.71) | -31.57 (27.05) | -30.73 (27.45) | -37.03 (26.66)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -33.24 (34.91) | -42.01 (28.18) | -29.57 (26.98) | -32.11 (27.54) | -38.47 (26.45)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -28.49 (34.27) | -38.03 (29.14) | -24.18 (28.11) | -28.51 (27.74) | -35.47 (27.47)

51. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: The number of participants who withdrew due to lack of efficacy up to week 12 was calculated.
Time Frame: Up to week 12
Population: Initial Randomization Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 101 | 104 | 102 | 200
Participants | 7 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.033, Fisher Exact — No Multiplicity Adjustment. Etanercept was open-label reference group and it was not included in statistical test
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.035, Fisher Exact — No Multiplicity Adjustment. Etanercept was open-label reference group and it was not included in statistical test

52. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 12
Description: The HAQ-DI (range 0 - 3) was composed of 20 items in 8 categories (Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, and Activities). Each category has at least two questions. Within each category, participants reported the amount of difficulty they have in performing the specific question items. Higher HAQ-DI score indicates greater disease activity.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | 0.03 (0.55) | -0.28 (0.55) | -0.37 (0.50) | -0.39 (0.48)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -0.34, 95% CI 2-sided [-0.48 to -0.20], Standard Error of Mean 0.07 — Based on analysis of covariance model: HAQ-DI Change = Treatment + Baseline HAQ-DI + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea., and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -0.40, 95% CI 2-sided [-0.53 to -0.26], Standard Error of Mean 0.07 — [estimate comment as in outcome 52, analysis 1]

53. Secondary Outcome: Change From Baseline in HAQ-DI Through Week 52
Description: as for outcome 52
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS, number of participants with available data at each study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 43 | 47 | 200
units on a scale
  Week 4: number analyzed (Participants) | 98 | 100 | 42 | 47 | 200
  Week 4 | -0.10 (0.35) | -0.19 (0.40) | -0.04 (0.32) | 0.01 (0.38) | -0.24 (0.43)
  Week 8: number analyzed (Participants) | 96 | 99 | 42 | 47 | 195
  Week 8 | -0.25 (0.48) | -0.31 (0.48) | -0.07 (0.45) | 0.02 (0.39) | -0.35 (0.45)
  Week 12: number analyzed (Participants) | 96 | 92 | 41 | 47 | 191
  Week 12 | -0.30 (0.55) | -0.38 (0.50) | -0.09 (0.55) | 0.03 (0.50) | -0.39 (0.47)
  Week 16: number analyzed (Participants) | 93 | 93 | 41 | 47 | 188
  Week 16 | -0.36 (0.58) | -0.41 (0.48) | -0.21 (0.49) | -0.12 (0.48) | -0.44 (0.50)
  Week 20: number analyzed (Participants) | 92 | 92 | 41 | 46 | 182
  Week 20 | -0.34 (0.56) | -0.46 (0.53) | -0.22 (0.58) | -0.21 (0.47) | -0.46 (0.52)
  Week 24: number analyzed (Participants) | 87 | 90 | 39 | 45 | 182
  Week 24 | -0.35 (0.58) | -0.46 (0.53) | -0.33 (0.59) | -0.26 (0.45) | -0.47 (0.53)
  Week 28: number analyzed (Participants) | 83 | 89 | 40 | 46 | 177
  Week 28 | -0.35 (0.58) | -0.49 (0.59) | -0.33 (0.53) | -0.23 (0.49) | -0.47 (0.51)
  Week 32: number analyzed (Participants) | 81 | 86 | 36 | 45 | 176
  Week 32 | -0.41 (0.56) | -0.50 (0.54) | -0.36 (0.54) | -0.29 (0.46) | -0.47 (0.56)
  Week 36: number analyzed (Participants) | 79 | 86 | 36 | 43 | 175
  Week 36 | -0.40 (0.56) | -0.50 (0.58) | -0.36 (0.51) | -0.25 (0.52) | -0.47 (0.55)
  Week 40: number analyzed (Participants) | 76 | 86 | 37 | 42 | 173
  Week 40 | -0.42 (0.60) | -0.51 (0.57) | -0.35 (0.50) | -0.28 (0.47) | -0.48 (0.54)
  Week 44: number analyzed (Participants) | 75 | 85 | 34 | 39 | 171
  Week 44 | -0.39 (0.58) | -0.51 (0.58) | -0.42 (0.63) | -0.27 (0.51) | -0.49 (0.55)
  Week 48: number analyzed (Participants) | 74 | 84 | 34 | 39 | 168
  Week 48 | -0.34 (0.56) | -0.52 (0.57) | -0.40 (0.59) | -0.31 (0.50) | -0.51 (0.53)
  Week 52: number analyzed (Participants) | 71 | 81 | 34 | 38 | 162
  Week 52 | -0.36 (0.57) | -0.54 (0.56) | -0.46 (0.57) | -0.29 (0.51) | -0.51 (0.53)
  EOT: number analyzed (Participants) | 102 | 101 | 42 | 47 | 200
  EOT | -0.30 (0.60) | -0.50 (0.57) | -0.37 (0.64) | -0.24 (0.50) | -0.47 (0.53)

54. Secondary Outcome: Change From Baseline in Short Form Health Survey - 36 Questions, Version 2 (SF-36v2) Physical Component Summary Score at Week 12
Description: The SF-36v2 was scored for the 8 subscales (each range: 0-100 scale): 1. physical functioning, 2. role physical, 3. bodily pain, 4. general health, 5. vitality, 6. social functioning, 7. role-emotional, and 8. mental health. Physical Component Summary Score, Mental Component Summary Score and Roll/Social Component Summary Score were calculated based on the 2007 General Japanese Population Means and Standard Deviations and coefficient. Component summary measures had means of 50 in 2007 General Japanese Population and deviation was expressed by the scale of 10. Higher score indicated better health state.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Peficitinib 100 m: Participants were assigned to receive peficitinib 100 mg/day for 52 weeks.
Arm/Group | Placebo | Peficitinib 100 m | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | 1.95 (12.20) | 8.36 (14.05) | 8.81 (10.54) | 8.53 (10.61)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 m; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = 6.87, 95% CI 2-sided [3.69 to 10.05], Standard Error of Mean 1.61 — Based on analysis of covariance model: SF-36v2 Change = Treatment + Baseline SF-36v2 + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = 6.98, 95% CI 2-sided [4.11 to 9.85], Standard Error of Mean 1.45 — [estimate comment as in outcome 54, analysis 1]

55. Secondary Outcome: Change From Baseline in SF-36v2 Physical Component Summary Score Through Week 52
Description: as for outcome 54
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: FAS, number of participants with available data at each study visit. The focus of data collection after Week 12 for participants transitioned from Placebo to Peficitinib was safety. Long term efficacy was not evaluated by the SF-36 questionnaire for them. These assessments were only conducted at Weeks 28 and 52 after transitioning to Peficitinib.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Etanercept: Participants were administered 50 mg of subcutaneous etanercept once weekly for 52 weeks.New Group 3 Description
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 200
  Week 4 | 3.82 (10.21) | 3.20 (10.49) | 6.10 (10.07)
  Week 8: number analyzed (Participants) | 96 | 99 | 195
  Week 8 | 6.43 (10.98) | 6.78 (9.99) | 7.35 (10.23)
  Week 12: number analyzed (Participants) | 96 | 92 | 191
  Week 12 | 9.93 (12.38) | 9.63 (10.33) | 8.40 (10.51)
  Week 28: number analyzed (Participants) | 83 | 89 | 177
  Week 28 | 10.85 (12.79) | 10.95 (12.04) | 10.28 (10.67)
  Week 52: number analyzed (Participants) | 71 | 81 | 162
  Week 52 | 13.07 (12.41) | 9.88 (12.51) | 11.18 (11.77)

56. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Summary Score at Week 12
Description: as for outcome 54
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | 0.00 (8.65) | 2.70 (7.59) | 3.69 (8.23) | 3.23 (8.24)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.004, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = 2.89, 95% CI 2-sided [0.91 to 4.87], Standard Error of Mean 1.00 — [estimate comment as in outcome 54, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = 3.25, 95% CI 2-sided [1.30 to 5.19], Standard Error of Mean 0.98 — [estimate comment as in outcome 54, analysis 1]

57. Secondary Outcome: Change From Baseline in SF-36v2 Mental Component Summary Score Through Week 52
Description: as for outcome 54
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
units on a scale
  Week 4: number analyzed (Participants) | 98 | 100 | 200
  Week 4 | 1.53 (7.19) | 1.72 (7.58) | 2.85 (8.07)
  Week 8: number analyzed (Participants) | 96 | 99 | 195
  Week 8 | 2.91 (7.39) | 3.55 (9.08) | 3.56 (8.49)
  Week 12: number analyzed (Participants) | 96 | 92 | 191
  Week 12 | 2.38 (7.53) | 4.01 (8.17) | 3.63 (7.95)
  Week 28: number analyzed (Participants) | 83 | 89 | 177
  Week 28 | 2.95 (8.07) | 3.52 (8.14) | 3.80 (7.66)
  Week 52: number analyzed (Participants) | 71 | 81 | 162
  Week 52 | 4.23 (8.17) | 4.39 (8.08) | 3.79 (8.38)

58. Secondary Outcome: Change From Baseline in SF-36v2 Role/Social Component Summary Score at Week 12
Description: as for outcome 54
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Units on a Scale | 0.17 (15.12) | 1.24 (14.40) | 7.04 (14.56) | 7.16 (13.23)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.210, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = 2.27, 95% CI 2-sided [-1.29 to 5.83], Standard Error of Mean 1.80 — [estimate comment as in outcome 54, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = 6.23, 95% CI 2-sided [2.74 to 9.71], Standard Error of Mean 1.77 — [estimate comment as in outcome 54, analysis 1]

59. Secondary Outcome: Change From Baseline in SF-36v2 Role/Social Component Summary Score Through Week 52
Description: as for outcome 54
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
Units on a Scale
  Week 4: number analyzed (Participants) | 98 | 100 | 200
  Week 4 | 0.40 (12.75) | 4.27 (12.02) | 4.06 (13.08)
  Week 8: number analyzed (Participants) | 96 | 99 | 195
  Week 8 | 3.80 (13.23) | 5.96 (14.60) | 6.51 (12.54)
  Week 12: number analyzed (Participants) | 96 | 92 | 191
  Week 12 | 1.68 (14.33) | 7.82 (14.66) | 7.49 (13.04)
  Week 28: number analyzed (Participants) | 83 | 89 | 177
  Week 28 | 4.18 (14.21) | 8.78 (14.20) | 7.31 (14.74)
  Week 52: number analyzed (Participants) | 71 | 81 | 162
  Week 52 | 3.88 (15.12) | 9.15 (13.39) | 8.36 (14.03)

60. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Percent Work Time Missed at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicate greater activity impairment. Multiply scores by 100 to express in percentages. Percent work time missed due to problem: Q2/(Q2+Q4).
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Percent Work Time
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 48 | 57 | 49 | 99
Percent Work Time | 6.78 (25.76) | -2.14 (18.47) | -6.80 (19.40) | -5.60 (20.63)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.027, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -8.55, 95% CI 2-sided [-16.11 to -1.00], Standard Error of Mean 3.81 — Based on analysis of covariance model: WPAI Change = Treatment + Baseline WPAI + the prior biologic-DMARD-IR (No, Yes) + concomitant DMARD use (No, Yes) + study region (Japan, Korea, and Taiwan)
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p = 0.010, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -10.17, 95% CI 2-sided [-17.88 to -2.47], Standard Error of Mean 3.88 — [estimate comment as in outcome 60, analysis 1]

61. Secondary Outcome: Change From Baseline in WPAI Percent Work Time Missed Through Week 52
Description: as for outcome 60
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: FAS, number of participants with available data at each study visit. The focus of data collection after Week 12 for participants transitioned from Placebo to Peficitinib was safety. Long term efficacy was not evaluated by the WPAI questionnaire for them. These assessments were only conducted at Weeks 28 and 52 after transitioning to Peficitinib.
Measure: Mean (Standard Deviation); unit: Percent Work Time
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
Percent Work Time
  Week 4: number analyzed (Participants) | 54 | 48 | 99
  Week 4 | -0.56 (20.13) | -6.35 (15.94) | -3.71 (17.34)
  Week 8: number analyzed (Participants) | 52 | 48 | 97
  Week 8 | -2.38 (16.15) | -6.10 (19.30) | -4.33 (15.57)
  Week 12: number analyzed (Participants) | 52 | 43 | 96
  Week 12 | -1.38 (18.13) | -6.69 (19.78) | -4.73 (18.54)
  Week 28: number analyzed (Participants) | 51 | 41 | 86
  Week 28 | -3.14 (24.48) | -6.46 (20.29) | -5.03 (18.18)
  Week 52: number analyzed (Participants) | 40 | 36 | 81
  Week 52 | -6.76 (22.20) | -6.35 (16.57) | -4.52 (14.91)

62. Secondary Outcome: Change From Baseline in WPAI Percent Impairment While Working at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicate greater activity impairment. Multiply scores by 100 to express in percentages. Percent impairment while working due to problem: Q5/10.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Percent Impairment
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 46 | 56 | 49 | 97
Percent Impairment | 4.13 (30.15) | -13.04 (30.45) | -16.12 (31.94) | -24.43 (25.82)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -20.67, 95% CI 2-sided [-30.44 to -10.89], Standard Error of Mean 4.92 — [estimate comment as in outcome 60, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -22.01, 95% CI 2-sided [-32.06 to -11.97], Standard Error of Mean 5.06 — [estimate comment as in outcome 60, analysis 1]

63. Secondary Outcome: Change From Baseline in WPAI Percent Impairment While Working Through Week 52
Description: as for outcome 62
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
percent impairment
  Week 4: number analyzed (Participants) | 53 | 48 | 96
  Week 4 | -6.42 (22.28) | -6.46 (27.48) | -18.33 (26.34)
  Week 8: number analyzed (Participants) | 51 | 48 | 96
  Week 8 | -14.31 (26.10) | -15.42 (27.75) | -20.52 (25.31)
  Week 12: number analyzed (Participants) | 51 | 43 | 95
  Week 12 | -13.33 (30.96) | -19.77 (31.66) | -24.11 (25.95)
  Week 28: number analyzed (Participants) | 49 | 41 | 86
  Week 28 | -17.35 (34.63) | -25.85 (28.10) | -29.53 (26.78)
  Week 52: number analyzed (Participants) | 38 | 36 | 81
  Week 52 | -20.79 (36.27) | -23.89 (30.55) | -31.36 (31.18)

64. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicate greater activity impairment. Multiply scores by 100 to express in percentages. Percent overall work impairment due to problem: Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)].
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Percent iImpairment
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 46 | 55 | 49 | 97
Percent iImpairment | 3.62 (30.49) | -12.20 (31.39) | -18.68 (33.81) | -24.68 (26.54)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -20.22, 95% CI 2-sided [-30.38 to -10.06], Standard Error of Mean 5.12 — [estimate comment as in outcome 60, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model; No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -23.67, 95% CI 2-sided [-34.16 to -13.17], Standard Error of Mean 5.28 — [estimate comment as in outcome 60, analysis 1]

65. Secondary Outcome: Change From Baseline in WPAI Percent Overall Work Impairment Through Week 52
Description: as for outcome 64
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Percent Impairment
Groups:
- Peficitinib 150 mg: assigned to receive peficitinib 150 mg/day for 52 weeks.
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
Percent Impairment
  Week 4: number analyzed (Participants) | 52 | 48 | 96
  Week 4 | -5.72 (21.61) | -8.67 (28.20) | -18.20 (26.96)
  Week 8: number analyzed (Participants) | 51 | 48 | 96
  Week 8 | -14.16 (27.22) | -17.44 (29.05) | -20.94 (25.88)
  Week 12: number analyzed (Participants) | 51 | 43 | 95
  Week 12 | -13.16 (32.11) | -22.84 (33.22) | -25.35 (26.68)
  Week 28: number analyzed (Participants) | 49 | 41 | 85
  Week 28 | -17.48 (34.87) | -28.68 (29.66) | -30.12 (28.21)
  Week 52: number analyzed (Participants) | 38 | 36 | 81
  Week 52 | -21.53 (35.95) | -24.75 (31.45) | -32.18 (31.81)

66. Secondary Outcome: Change From Baseline in WPAI Percent Activity Impairment at Week 12
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to the rheumatoid arthritis; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the rheumatoid arthritis on productivity while working; Q6=Impact of the rheumatoid arthritis on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicate greater activity impairment. Multiply scores by 100 to express in percentages. Percent activity impairment due to problem: Q6/10.
Time Frame: Baseline and Week 12/ET
Population: FAS, number of participants with both baseline and available post-baseline data up to week 12. LOCF was used.
Measure: Mean (Standard Deviation); unit: Percent Impairment
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 99 | 102 | 101 | 200
Percent Impairment | -4.65 (26.39) | -19.61 (29.62) | -24.65 (28.27) | -26.40 (24.50)
Statistical Analysis 1: Comparison: Placebo vs Peficitinib 100 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -17.30, 95% CI 2-sided [-24.00 to -10.61], Standard Error of Mean 3.39 — [estimate comment as in outcome 60, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Peficitinib 150 mg; Treatment Difference vs Placebo; Test type: Superiority; p < 0.001, Covariance model — No multiplicity adjustment. Etanercept was open-label reference group and it was not included in statistical test; LS mean = -20.41, 95% CI 2-sided [-26.59 to -14.24], Standard Error of Mean 3.13 — [estimate comment as in outcome 60, analysis 1]

67. Secondary Outcome: Change From Baseline in WPAI Percent Activity Impairment Through Week 52
Description: as for outcome 66
Time Frame: Baseline and Week 4, 8, 12, 28, and 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 104 | 102 | 200
percent impairment
  Week 4: number analyzed (Participants) | 98 | 100 | 200
  Week 4 | -10.92 (24.75) | -11.30 (21.82) | -17.90 (23.11)
  Week 8: number analyzed (Participants) | 96 | 99 | 195
  Week 8 | -20.10 (26.89) | -23.64 (26.05) | -25.33 (23.95)
  Week 12: number analyzed (Participants) | 95 | 92 | 191
  Week 12 | -21.47 (29.53) | -26.74 (28.48) | -27.33 (23.90)
  Week 28: number analyzed (Participants) | 83 | 89 | 177
  Week 28 | -25.18 (31.40) | -30.00 (27.80) | -30.34 (26.86)
  Week 52: number analyzed (Participants) | 71 | 81 | 162
  Week 52 | -28.17 (30.01) | -34.07 (27.69) | -31.79 (26.96)

68. Secondary Outcome: Number of Participants With Adverse Events During the First 12 Weeks
Description: Treatment-emergent adverse events (TEAEs) were defined as any AE that started or worsened in severity after initial dose of study drug or reference drug through week 52 or withdrawal. TEAEs were summarized using MedDRA (Version 11.1) by System Organ Class (SOC) and Preferred Term (PT). Participants reporting more than 1 AE for a given MedDRA PT were counted only once for that term. Participants reporting more than 1 AE within a SOC were counted only once for the SOC total. Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade: grade 3 = severe or medically significant, grade 4 = life threatening, grade 5 = death related to AE.
Time Frame: Week 0 to Week 12
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Peficitinib 100 mg | Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 101 | 104 | 102 | 200
Participants
  TEAEs | 54 | 49 | 55 | 119
  Drug-related TEAEs | 29 | 33 | 38 | 75
  TEAEs leading to death | 0 | 0 | 0 | 0
  Serious TEAEs | 4 | 3 | 2 | 4
  Drug-related serious TEAEs | 3 | 2 | 1 | 4
  ≥ Grade 3 TEAEs | 8 | 6 | 3 | 6
  TEAEs leading to discontinuation | 4 | 6 | 3 | 5
  Drug-related TEAEs leading to discontinuation | 1 | 4 | 2 | 5
  Serious TEAEs leading to discontinuation | 2 | 2 | 2 | 2
  Drug-related serious TEAEs leading to discont. | 1 | 1 | 1 | 2

69. Secondary Outcome: Number of Participants With Adverse Events From Week 12
Description: Treatment-emergent adverse events (TEAEs) were defined as any AE that started or worsened in severity after initial dose of study drug or reference drug through week 52 or withdrawal. TEAEs were summarized using MedDRA (Version 11.1) by SOC and PT. Participants reporting more than 1 AE for a given MedDRA PT were counted only once for that term. Participants reporting more than 1 AE within a SOC were counted only once for the SOC total. Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade: grade 3 = severe or medically significant, grade 4 = life threatening, grade 5 = death related to AE.
Time Frame: Week 12 to week 52, plus 28 days after the week 52 visit for participants who did not enroll in the extension study
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Peficitinib 100 mg | Peficitinib 150 mg | Placebo / Peficitinib 100 mg | Placebo / Peficitinib 150 mg | Etanercept
Number analyzed (Participants) | 96 | 93 | 43 | 47 | 191
Participants
  TEAEs | 78 | 79 | 41 | 37 | 156
  Drug-related TEAEs | 50 | 47 | 27 | 26 | 93
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 5 | 6 | 4 | 5 | 14
  Drug-related serious TEAEs | 2 | 2 | 2 | 2 | 5
  ≥ Grade 3 TEAEs | 9 | 16 | 2 | 12 | 23
  TEAEs leading to discontinuation | 7 | 3 | 2 | 4 | 8
  Drug-related TEAEs leading to discontinuation | 3 | 2 | 2 | 4 | 6
  Serious TEAEs leading to discontinuation | 4 | 0 | 1 | 2 | 3
  Drug-related serious TEAEs leading to discont. | 2 | 0 | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Week 0 to week 12, and from week 12 to week 52, plus 28 days after the week 52 visit for participants who did not enroll in the extension study.
Description: The safety analysis set (SAF) consisted of all participants who received at least one dose of study drugs.
Groups:
- Weeks 0-12: Placebo: Participants were assigned to receive placebo to peficitinib once a day until week 12.
- Weeks 0-12: Peficitinib 100 mg: Participants were assigned to receive peficitinib 100 mg/day until 12 weeks.
- Weeks 0-12: Peficitinib 150 mg: Participants were assigned to receive peficitinib 150 mg/day until 12 weeks.
- Weeks 0-12: Etanercept: Participants were administered 50 mg of subcutaneous etanercept once weekly until 12 weeks.
- Weeks 12-52: Peficitinib 100 mg: Participants were assigned to receive peficitinib 100 mg/day until 12 weeks and from week 12 to week 52.
- Weeks 12-52: Peficitinib 150 mg: Participants were assigned to receive peficitinib 150 mg/day until 12 weeks and from week 12 to week 52.
- Weeks 12-52: Placebo / Peficitinib 100 mg: Participants were assigned to receive placebo to peficitinib once a day until week 12 and peficitinib 100 mg/day from week 12 to week 52.
- Weeks 12-52: Placebo / Peficitinib 150 mg: Participants were assigned to receive placebo to peficitinib once a day until week 12 and peficitinib 150 mg/day from week 12 to week 52.
- Weeks 12-52: Etanercept: Participants were administered 50 mg of subcutaneous etanercept once weekly until 12 weeks and from week 12 to week 52.
Arm/Group | Weeks 0-12: Placebo | Weeks 0-12: Peficitinib 100 mg | Weeks 0-12: Peficitinib 150 mg | Weeks 0-12: Etanercept | Weeks 12-52: Peficitinib 100 mg | Weeks 12-52: Peficitinib 150 mg | Weeks 12-52: Placebo / Peficitinib 100 mg | Weeks 12-52: Placebo / Peficitinib 150 mg | Weeks 12-52: Etanercept
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/104 | 0/102 | 0/200 | 0/96 | 0/93 | 0/43 | 0/47 | 0/191
Serious Adverse Events (participants affected / at risk) | 4/101 | 3/104 | 2/102 | 4/200 | 5/96 | 6/93 | 4/43 | 5/47 | 14/191
Other Adverse Events (participants affected / at risk) | 27/101 | 30/104 | 39/102 | 63/200 | 50/96 | 42/93 | 28/43 | 23/47 | 94/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weeks 0-12: Placebo (N=101) | Weeks 0-12: Peficitinib 100 mg (N=104) | Weeks 0-12: Peficitinib 150 mg (N=102) | Weeks 0-12: Etanercept (N=200) | Weeks 12-52: Peficitinib 100 mg (N=96) | Weeks 12-52: Peficitinib 150 mg (N=93) | Weeks 12-52: Placebo / Peficitinib 100 mg (N=43) | Weeks 12-52: Placebo / Peficitinib 150 mg (N=47) | Weeks 12-52: Etanercept (N=191)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Social stay hospitalisation (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weeks 0-12: Placebo (N=101) | Weeks 0-12: Peficitinib 100 mg (N=104) | Weeks 0-12: Peficitinib 150 mg (N=102) | Weeks 0-12: Etanercept (N=200) | Weeks 12-52: Peficitinib 100 mg (N=96) | Weeks 12-52: Peficitinib 150 mg (N=93) | Weeks 12-52: Placebo / Peficitinib 100 mg (N=43) | Weeks 12-52: Placebo / Peficitinib 150 mg (N=47) | Weeks 12-52: Etanercept (N=191)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 3 (4)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 25 (77) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (63)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 0 (0) | 7 (7) | 9 (9) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 5 (5) | 7 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 5 (5)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 4 (4) | 1 (1) | 3 (6)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 5 (5) | 2 (2) | 2 (2) | 8 (8)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (11) | 19 (19) | 16 (17) | 21 (30) | 15 (21) | 13 (18) | 8 (11) | 49 (77)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 7 (11) | 3 (4) | 0 (0) | 4 (4) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (4) | 3 (3) | 3 (3) | 4 (5) | 4 (4) | 5 (7) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 6 (9) | 7 (7) | 3 (3) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 (17) | 2 (3) | 2 (12) | 3 (4) | 3 (3) | 3 (3) | 2 (3) | 0 (0) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 4 (5) | 1 (1) | 3 (3) | 8 (8)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (4) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 9 (10)

LIMITATIONS AND CAVEATS:
The focus of data collection after Week 12 for participants who transitioned from Placebo to Peficitinib was safety. Efficacy was not evaluated by the SF-36 and WPAI questionnaire after Week 12 for participants first assigned to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02308163/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02308163/SAP_001.pdf